CLINICAL TRIAL: NCT00265317
Title: Randomized, Double-Blind, Phase 2 Study Of Erlotinib With Or Without SU011248 In The Treatment Of Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study In Patients With Non-Small Cell Lung Cancer Testing If Erlotinib Plus SU011248 (Sunitinib) Is Better Than Erlotinib Alone
Acronym: SUN1058
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6181058
Record Dates: First submitted 2005-12-12; First posted 2005-12-14 (Estimated); Results first posted 2011-06-10 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-small cell lung cancer; sunitinib; erlotinib; Phase 2
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Sunitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: erlotinib; Drug: sunitinib
- B (Active Comparator)
  Interventions: Drug: erlotinib; Drug: placebo

INTERVENTIONS:
Drug: erlotinib — erlotinib 150 mg daily by tablets in a continuous regimen, until progression or unacceptable toxicity
  Arms: A
Drug: sunitinib — Sunitinib 37.5 mg daily by oral capsule in a continuous regimen plus erlotinib 150 mg daily by tablets in a continuous regimen, until progression or unacceptable toxicity
  Other Names: Sutent
  Arms: A
Drug: erlotinib — erlotinib 150 mg daily by tablets in a continuous regimen, until progression or unacceptable toxicity
  Arms: B
Drug: placebo — Placebo daily by oral capsule in a continuous regimen plus erlotinib 150 mg daily by tablets in a continuous regimen, until progression or unacceptable toxicity
  Arms: B

SUMMARY:
This study will test whether treatment with erlotinib plus SU011248 is better than erlotinib alone in patients with advanced/metastatic lung cancer who have received previous treatment with a platinum-based regimen

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced/metastatic non-small cell lung cancer
* Prior treatment with no more than 2 chemotherapy regimens including a platinum-based regimen

Exclusion Criteria:

* Prior treatment with any receptor tyrosine kinase inhibitors, Vascular endothelial growth factor (VEGF) inhibitors or other angiogenic inhibitors
* History of or known brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2006-06; Primary Completion 2010-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (30):
- United States (16):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Antioch, California
  - Pfizer Investigational Site, Palm Springs, California
  - Pfizer Investigational Site, Pleasant Hill, California
  - Pfizer Investigational Site, San Leandro, California
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, City of Saint Peters, Missouri
  - Pfizer Investigational Site, Creve Coeur, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Chapel Hill, North Carolina
  - Pfizer Investigational Site, Clinton, North Carolina
  - Pfizer Investigational Site, Goldsboro, North Carolina
  - Pfizer Investigational Site, Wilson, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Houston, Texas
- Canada (2):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Hamilton, Ontario
- Hungary (2):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Törökbálint
- Italy (2):
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Monteforte Irpino, AV
- Netherlands (2):
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Groningen
- Poland (2):
  - Pfizer Investigational Site, Bydgoszcz
  - Pfizer Investigational Site, Gdansk
- Romania (3):
  - Pfizer Investigational Site, Cluj-Napoca, Cluj
  - Pfizer Investigational Site, Bucharest, Sector 2
  - Pfizer Investigational Site, Bucharest
- Pfizer Investigational Site, Santander, Cantabria, Spain

REFERENCES:
- [Derived] Groen HJ, Socinski MA, Grossi F, Juhasz E, Gridelli C, Baas P, Butts CA, Chmielowska E, Usari T, Selaru P, Harmon C, Williams JA, Gao F, Tye L, Chao RC, Blumenschein GR Jr. A randomized, double-blind, phase II study of erlotinib with or without sunitinib for the second-line treatment of metastatic non-small-cell lung cancer (NSCLC). Ann Oncol. 2013 Sep;24(9):2382-9. doi: 10.1093/annonc/mdt212. Epub 2013 Jun 20. PMID 23788751
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181058&StudyName=A%20Study%20In%20Patients%20With%20Non-Small%20Cell%20Lung%20Cancer%20Testing%20If%20Erlotinib%20Plus%20SU011248%20%28sunitinib%29%20Is%20Better%20Than%20Erlotinib%20Alone

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib + Erlotinib (Original Lead-In): Sunitinib 37.5 mg oral capsules once daily (QD) for 28 days each cycle with exception of Cycle 2 (27 days) and Erlotinib 150 mg oral tablets QD for 28 days each cycle with exception of Cycle 1 (35 days).
- Sunitinib + Erlotinib (Amended Lead-in): Sunitinib 37.5 mg oral capsules QD for 28 days each cycle (27 days in Cycle 1, Arm A or 13 days in Cycle 1, Arm B) and Erlotinib 150 mg oral tablets QD for 28 days each cycle (7 days in Cycle 1, Arm A or 26 days in Cycle 1, Arm B)
- Sunitinib + Erlotinib: Sunitinib oral capsules, 37.5 mg QD in a continuous regimen, expressed in 4-week cycles and Erlotinib 150 mg oral tablets QD in a continuous regimen expressed in 4-week cycles.
- Erlotinib + Placebo: Erlotinib 150 mg oral tablets QD in a continuous regimen expressed in 4-week cycles and Placebo oral capsules QD in a continuous regimen expressed in 4-week cycles.
Period: Lead-In
Arm/Group | Sunitinib + Erlotinib (Original Lead-In) | Sunitinib + Erlotinib (Amended Lead-in) | Sunitinib + Erlotinib | Erlotinib + Placebo
Started | 13 | 17 | 0 | 0
Completed | 1 | 0 | 0 | 0
Not Completed | 12 | 17 | 0 | 0
Not completed — Objective progression or relapse | 6 | 11 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 0 | 0
Not completed — Death | 3 | 5 | 0 | 0
Not completed — Withdrawal/other than adverse event | 1 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Sunitinib + Erlotinib (Original Lead-In) | Sunitinib + Erlotinib (Amended Lead-in) | Sunitinib + Erlotinib | Erlotinib + Placebo
Started | 0 | 0 | 65 | 67
Completed | 0 | 0 | 1 | 2
Not Completed | 0 | 0 | 64 | 65
Not completed — Objective progression or relapse | 0 | 0 | 37 | 38
Not completed — Global deterioration of health status | 0 | 0 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 7 | 5
Not completed — Death | 0 | 0 | 12 | 15
Not completed — Protocol Violation | 0 | 0 | 1 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal/other than adverse event | 0 | 0 | 2 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sunitinib + Erlotinib (Original Lead-In) | Sunitinib + Erlotinib (Amended Lead-in) | Sunitinib + Erlotinib | Erlotinib + Placebo | Total
Number analyzed (Participants) | 13 | 17 | 65 | 67 | 162
Age, Customized [Number; unit: participants]
  Less than 65 years | 7 | 10 | 47 | 43 | 107
  Greater than or equal to 65 years | 6 | 7 | 17 | 24 | 54
  Unknown or Not Collected | 0 | 0 | 1 | 0 | 1
Sex/Gender, Customized [Number; unit: participants]
  Female | 6 | 6 | 25 | 22 | 59
  Male | 7 | 11 | 39 | 45 | 102
  Unknown or Not Collected | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS=time from randomization date to date of first documentation of progressive disease (PD; defined as greater than or equal to [≥]20% increase in sum of longest dimensions of target lesions taking as a reference smallest sum of longest dimensions recorded since first dose or appearance of ≥1 new lesions) or death on-study due to any cause, whichever occurred first based on third party independent imaging review laboratory assessment. PFS calculated as (first event date minus randomization date plus 1) divided by 7.02. Used 7.02 days as it equals 365 days per year divided by 52 weeks per year.
Time Frame: From randomization to Weeks 8 and 12, then every 8 weeks until disease progression or death (up to Month 17)
Population: Full Analysis Set (FA):all participants in randomized phase randomized with study medication assignment designated according to initial randomization, regardless of whether participants actually received study medication or received different medication from what they were randomized.
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- Sunitinib + Erlotinib: Erlotinib 150 mg oral tablets once daily (QD) in a continuous regimen expressed in 4-week cycles and Sunitinib 37.5 mg oral capsules QD in a continuous regimen expressed in 4-week cycles.
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Weeks | 12.3 [8.10 to 19.50] | 8.5 [8.00 to 12.30]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Sample size for randomized portion of study determined based on these assumptions: median PFS (erlotinib)=10 weeks, accrual time=12 months. With 6 months follow-up, study was powered to detect a difference in PFS of 5 weeks. 1-sided log rank test comparing the 2 treatment groups with 115 events of PD or death among a target sample size of 126 participants (63 per group) achieved 80% power at a 10% significance level to detect a 50% improvement in PFS from 10 to 15 weeks; Test type: Superiority or Other; p = 0.3206, Log Rank — Primary analysis was based on an unstratified 1-sided log rank test with alpha=0.1; Hazard Ratio (HR) = 0.898, 80% CI 2-sided [0.575 to 1.404]

2. Secondary Outcome: Percentage of Participants With Objective Response
Description: Objective Response Rate (ORR)=participants with confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST,Version 1.0) based on third party independent imaging review laboratory assessment. A CR was defined as the disappearance of all target lesions that persisted on repeat imaging study at least 4 weeks after initial documentation of response. A PR was defined as a ≥30% decrease in sum of longest dimensions of target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: From randomization to Weeks 8 and 12, then every 8 weeks until disease progression or death (up to Month 17)
Population: FA Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Percentage of Participants | 4.62 [0.96 to 12.90] | 2.99 [0.36 to 10.37]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; 95% confidence interval (CI) calculated based on f-distribution; Test type: Superiority or Other; p = 0.6251, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.546, 95% CI 2-sided [0.267 to 8.954]

3. Secondary Outcome: Time to Tumor Progression (TTP)
Description: TTP was defined as the time from date of randomization to first documentation of PD based on third party independent imaging review laboratory assessment. TTP was calculated as (first event date minus randomization date plus 1) divided by 7.02.
Time Frame: From randomization to Weeks 8 and 12, then every 8 weeks until disease progression or death (up to Month 17)
Population: FA Set
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Weeks | 12.3 [8.80 to 20.10] | 10.1 [8.10 to 13.00]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Test type: Superiority or Other; p = 0.3732, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.921, 95% CI 2-sided [0.572 to 1.485]

4. Secondary Outcome: Duration of Response (DR)
Description: DR was defined as time from first documentation of objective tumor response (CR or PR) that was subsequently confirmed to the first documentation of PD or death on-study due to any cause, whichever occurred first. DR was calculated as (first date of PD or death minus first date of CR or PR that was subsequently confirmed plus 1) divided by 7.02.
Time Frame: From randomization to Weeks 8 and 12, then every 8 weeks until disease progression or death (up to Month 17)
Population: FA subset of participants with a confirmed objective response were to be analyzed. As only 3 and 2 responses were observed, duration of response was not analyzed.
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as time from date of randomization to date of death due to any cause. OS was calculated as (date of death minus date of randomization plus 1) divided by 30.4. For participants still alive at the time of analysis, OS time was censored on last date that participants were known to be alive.
Time Frame: From randomization until death (up to Month 17)
Population: FA Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Months | 8.2 [5.70 to 11.30] | 7.6 [5.30 to 13.40]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Test type: Superiority or Other; p = 0.6171, Log Rank — p-value from 1-sided unstratified log-rank test; Hazard Ratio (HR) = 1.066, 95% CI 2-sided [0.705 to 1.612]

6. Secondary Outcome: Percentage of Participants Surviving at 1 Year
Description: Percentage of participants alive at 1 year after date of first administration of study medication.
Time Frame: From randomization until death (up until Month 17)
Population: FA Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Percentage of Participants | 32 [0.197 to 0.443] | 42 [0.301 to 0.542]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib; Percentage of participants surviving at 1 year in the Sunitinib + Erlotinib Treatment Group, estimated using the Kaplan-Meier method; Test type: Superiority or Other; Percentage = 32, 95% CI 2-sided [19.7 to 44.3]
Statistical Analysis 2: Comparison: Erlotinib + Placebo; Percentage of participants surviving at 1 year in the Erlotinib + Placebo Treatment Group, estimated using the Kaplan-Meier method; Test type: Superiority or Other; Percentage = 42, 95% CI 2-sided [30.1 to 54.2]

7. Secondary Outcome: Area Under the Curve From Time Zero to 24 Hours [AUC(0-24)] of Erlotinib
Description: AUC0-24=Area under the plasma concentration versus time curve from time zero (pre-dose) to 24 hours (0-24) of erlotinib
Time Frame: Days 1 and 22 (Cycle 1) at 0, 1, 2, 4, 6, 8, and 24 hours postdose
Population: Amended Lead-in Cohort Arm A: participants received sunitinib QD for 28 days each cycle (27 days in Cycle 1) and erlotinib QD for 28 days each cycle (7 days in Cycle 1)
Measure: Mean (Standard Deviation); unit: micrograms (mcg)*hour(hr)/milliliter (mL
Groups:
- Sunitinib + Erlotinib (Amended Lead-In Arm A): Sunitinib 37.5 mg oral capsules QD for 28 days each cycle (27 days in Cycle 1) and Erlotinib 150 mg oral tablets QD for 28 days each cycle (7 days in Cycle 1).
Arm/Group | Sunitinib + Erlotinib (Amended Lead-In Arm A)
Number analyzed (Participants) | 7
micrograms (mcg)*hour(hr)/milliliter (mL
  Cycle 1, Day 1 | 12.96 (4.00)
  Cycle 1, Day 22 | 11.87 (4.35)

8. Secondary Outcome: AUC(0-24) of Sunitinib
Description: AUC0-24=Area under the plasma concentration versus time curve from time zero (pre-dose) to 24 hours (0-24) of sunitinib
Time Frame: Days 1 and 15 of Cycle 1 at 0, 1, 2, 4, 6, 8, and 24 hours postdose
Population: Amended Lead-In Cohort Arm B: participants received sunitinib for 28 days each cycle (13 days in Cycle 1) and erlotinib QD for 28 days each cycle (26 days in Cycle 1).
Measure: Mean (Standard Deviation); unit: nanograms (ng)*hr/mL
Groups:
- Sunitinib+Erlotinib (Amended Lead-In Arm B): Sunitinib 37.5 mg oral capsules QD for 28 days each cycle (13 days in Cycle 1) and Erlotinib 150 mg oral tablets QD for 28 days each cycle (26 days in Cycle 1)
Arm/Group | Sunitinib+Erlotinib (Amended Lead-In Arm B)
Number analyzed (Participants) | 8
nanograms (ng)*hr/mL
  Cycle 1, Day 1 | 372.76 (105.21)
  Cycle 1, Day 15 | 231.61 (69.42)

9. Secondary Outcome: AUC(0-24) of SU-012662 (Metabolite of Sunitinib)
Description: AUC0-24=Area under the plasma concentration versus time curve from time zero (pre-dose) to 24 hours (0-24) of SU-012662 (metabolite of sunitinib)
Time Frame: Days 1 and 15 of Cycle 1 at 0, 1, 2, 4, 6, 8, and 24 hours postdose
Population: Amended Lead-In Cohort Arm B
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Sunitinib+Erlotinib (Amended Lead-In Arm B)
Number analyzed (Participants) | 8
ng*hr/mL
  Cycle 1, Day 1 | 50.06 (22.76)
  Cycle 1, Day 15 | 99.57 (39.48)

10. Secondary Outcome: AUC(0-24) of Total Drug (Sunitinib + SU-012662)
Description: AUC0-24=Area under the plasma concentration versus time curve from time zero (pre-dose) to 24 hours (0-24) of total drug (sunitinib + SU-012662)
Time Frame: Days 1 and 15 of Cycle 1 at 0, 1, 2, 4, 6, 8, and 24 hours postdose
Population: Amended Lead-In Cohort Arm B
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Sunitinib+Erlotinib (Amended Lead-In Arm B)
Number analyzed (Participants) | 8
ng*hr/mL
  Cycle 1, Day 1 | 422.93 (123.29)
  Cycle 1, Day 15 | 331.45 (88.67)

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Erlotinib
Time Frame: Days 1 and 22 (Cycle 1) at 0, 1, 2, 4, 6, 8, and 24 hours postdose
Population: Amended Lead-In Cohort Arm A
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Sunitinib + Erlotinib (Amended Lead-In Arm A)
Number analyzed (Participants) | 7
mcg/mL
  Cycle 1, Day 1 | 0.99 (0.48)
  Cycle 1, Day 22 | 0.86 (0.37)

12. Secondary Outcome: Cmax of Sunitinib
Time Frame: Days 1 and 15 of Cycle 1 at 0, 1, 2, 4, 6, 8, 24 and 48 hours postdose
Population: Amended Lead-In Cohort Arm B
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib+Erlotinib (Amended Lead-In Arm B)
Number analyzed (Participants) | 8
ng/mL
  Cycle 1, Day 1 | 21.61 (6.76)
  Cycle 1, Day 15 | 13.59 (5.88)

13. Secondary Outcome: Cmax of SU-012662 (Metabolite of Sunitinib)
Time Frame: Days 1 and 15 of Cycle 1 at 0, 1, 2, 4, 6, 8, 24 and 48 hours postdose
Population: Amended Lead-In Cohort Arm B
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib+Erlotinib (Amended Lead-In Arm B)
Number analyzed (Participants) | 8
ng/mL
  Cycle 1, Day 1 | 3.09 (1.33)
  Cycle 1, Day 15 | 6.83 (4.22)

14. Secondary Outcome: Cmax of Total Drug (Sunitinib + SU-012662)
Time Frame: Days 1 and 15 of Cycle 1 at 0, 1, 2, 4, 6, 8, 24 and 48 hours postdose
Population: Amended Lead-In Cohort Arm B
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib+Erlotinib (Amended Lead-In Arm B)
Number analyzed (Participants) | 8
ng/mL
  Cycle 1, Day 1 | 24.51 (7.72)
  Cycle 1, Day 15 | 20.09 (7.80)

15. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC0-inf) for Erlotinib
Description: AUC (0-inf) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf) for erlotinib. It is obtained from AUC from time zero (pre-dose) to last quantifiable concentration(AUC[0-t]) plus AUC from time last quantifiable concentration extrapolated infinite time (AUC[t-inf])
Time Frame: Days 1 and 22 (Cycle 1) at 0, 1, 2, 4, 6, 8, and 24 hours postdose; predose on Days 22 and 23 (Cycle 1)
Population: Amended Lead-In Cohort Arm A; Due to the long half-life of the drug and sample collection just up to 24 hours only, AUC(0-inf) could not be accurately estimated.
Arm/Group | Sunitinib + Erlotinib (Amended Lead-In Arm A)
Number analyzed (Participants) | 0

16. Secondary Outcome: AUC(0-inf) for Sunitinib
Description: AUC (0 - inf) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf) for sunitinib. It is obtained from AUC(0-t) plus AUC(t-inf)
Time Frame: Days 1 and 15 of Cycle 1 at 0, 1, 2, 4, 6, 8, 24 and 48 hours postdose; predose on Days 15, 16, and 17 (Cycle 1)
Population: Amended Lead-In Cohort Arm B; Due to the long half-life of the drug and sample collection just up to 48 hours only, AUC(0-inf) could not be accurately estimated.
Groups:
- Sunitinib + Erlotinib (Amended Lead-In Arm B): Sunitinib 37.5 mg oral capsules QD for 28 days each cycle (13 days in Cycle 1) and Erlotinib 150 mg oral tablets QD for 28 days each cycle (26 days in Cycle 1)
Arm/Group | Sunitinib + Erlotinib (Amended Lead-In Arm B)
Number analyzed (Participants) | 0

17. Secondary Outcome: AUC(0-inf) for SU-012662 (Metabolite of Sunitinib)
Description: AUC(0-inf) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf) for SU-012662 (metabolite of sunitinib). It is obtained from AUC(0-t) plus AUC(t-inf)
Time Frame: Days 1 and 15 of Cycle 1 at 0, 1, 2, 4, 6, 8, 24 and 48 hours postdose; predose on Days 15, 16, and 17 (Cycle 1)
Population: as for outcome 16
Arm/Group | Sunitinib + Erlotinib (Amended Lead-In Arm B)
Number analyzed (Participants) | 0

18. Secondary Outcome: AUC(0-inf) for Total Drug (Sunitinib + SU-012662)
Description: AUC(0-inf) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf) for total drug (sunitinib + SU-012662). It is obtained from AUC(0-t) plus AUC(t-inf)
Time Frame: Days 1 and 15 of Cycle 1 at 0, 1, 2, 4, 6, 8, 24 and 48 hours postdose; predose on Days 15, 16, and 17 (Cycle 1)
Population: as for outcome 16
Arm/Group | Sunitinib + Erlotinib (Amended Lead-In Arm B)
Number analyzed (Participants) | 0

19. Secondary Outcome: Plasma Decay Half-life (t1/2) of Erlotinib
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Days 1 and 22 (Cycle 1) at 0, 1, 2, 4, 6, 8, and 24 hours postdose
Population: Amended Lead-In Cohort Arm A; Due to the long half-life of the drug and sample collection just up to 24 hours only, t1/2 could not be accurately estimated.
Arm/Group | Sunitinib + Erlotinib (Amended Lead-In Arm A)
Number analyzed (Participants) | 0

20. Secondary Outcome: Plasma Decay Half-life (t1/2) of Sunitinib
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Days 1 and 15 of Cycle 1 at 0, 1, 2, 4, 6, 8, 24 and 48 hours postdose
Population: Amended Lead-In Cohort Arm B; Due to the long half-life of the drug and sample collection just up to 48 hours only, t1/2 could not be accurately estimated.
Arm/Group | Sunitinib + Erlotinib (Amended Lead-In Arm B)
Number analyzed (Participants) | 0

21. Secondary Outcome: Erlotinib Clearance at Steady State After Oral Administration (CL/F)
Time Frame: Day 15 (Cycle 1) at 0, 1, 2, 4, 6, 8, and 24 hours postdose
Population: Number of participants with calculable data in Original Lead-In; after protocol amendment 3, the study design was modified (steady-state versus single dose), due to the long half-life of the drug, sample collection just up to 24 hours was not sufficient for the calculation of CL/F for Amended Lead-In Arm A.
Measure: Mean (Standard Deviation); unit: Liters (L)/hr
Groups:
- Sunitinib + Erlotinib (Original Lead-In); Sunitinib + Erlotinib (Amended Lead-In Arm A): Sunitinib 37.5 mg oral capsules QD for 28 days each cycle (27 days in Cycle 1) and Erlotinib 150 mg oral tablets QD for 28 days each cycle (7 days in Cycle 1).
Arm/Group | Sunitinib + Erlotinib (Original Lead-In) | Sunitinib + Erlotinib (Amended Lead-In Arm A)
Number analyzed (Participants) | 8 | 0
Liters (L)/hr | 5.52 (3.65) |

22. Secondary Outcome: Sunitinib Clearance at Steady State After Oral Administration (CL/F)
Time Frame: Day 15 of Cycle 1 at 0, 1, 2, 4, 6, 8, 24 and 48 hours postdose
Population: Number of participants with calculable data in Original Lead-In Cohort; after protocol amendment 3, the study design was modified (steady-state versus single dose), due to the long half-life of the drug, sample collection just up to 48 hours was not sufficient for the calculation of CL/F for Amended Lead-In Arm B.
Measure: Mean (Standard Deviation); unit: L/hr
Groups:
- Sunitinib + Erlotinib (Original Lead-In): Sunitinib 37.5 mg oral capsules once daily (QD) for 28 days each cycle with exception of Cycle 2 (27 days)and Erlotinib 150 mg oral tablets QD for 28 days each cycle with exception of Cycle 1 (35 days).
Arm/Group | Sunitinib + Erlotinib (Original Lead-In) | Sunitinib + Erlotinib (Amended Lead-In Arm B)
Number analyzed (Participants) | 8 | 0
L/hr | 63.28 (13.50) |

23. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for Erlotinib
Time Frame: Days 1 and 22 (Cycle 1) at 0, 1, 2, 4, 6, 8, and 24 hours postdose
Population: Amended Lead-In Cohort Arm A
Measure: Median (Full Range); unit: Hours
Arm/Group | Sunitinib + Erlotinib (Amended Lead-In Arm A)
Number analyzed (Participants) | 8
Hours
  Cycle 1, Day 1 | 2.00 [1.00 to 6.00]
  Cycle 1, Day 22 | 2.00 [1.00 to 24.00]

24. Secondary Outcome: Tmax for Sunitinib
Time Frame: Days 1 and 15 of Cycle 1 at 0, 1, 2, 4, 6, 8, 24 and 48 hours postdose
Population: Amended Lead-In Cohort Arm B
Measure: Median (Full Range); unit: Hours
Arm/Group | Sunitinib + Erlotinib (Amended Lead-In Arm B)
Number analyzed (Participants) | 8
Hours
  Cycle 1, Day 1 | 6.00 [4.00 to 8.00]
  Cycle 1, Day 15 | 6.00 [4.00 to 24.00]

25. Secondary Outcome: Tmax for SU-012662 (Metabolite of Sunitinib)
Time Frame: Days 1 and 15 of Cycle 1 at 0, 1, 2, 4, 6, 8, 24 and 48 hours postdose
Population: Amended Lead-In Cohort Arm B
Measure: Median (Full Range); unit: Hours
Arm/Group | Sunitinib + Erlotinib (Amended Lead-In Arm B)
Number analyzed (Participants) | 8
Hours
  Cycle 1, Day 1 | 4.00 [2.00 to 48.00]
  Cycle 1, Day 15 | 4.00 [4.00 to 8.00]

26. Secondary Outcome: Tmax for Total Drug (Sunitinib + SU-012662)
Time Frame: Days 1 and 15 of Cycle 1 at 0, 1, 2, 4, 6, 8, 24 and 48 hours postdose
Population: Amended Lead-In Cohort Arm B
Measure: Median (Full Range); unit: Hours
Arm/Group | Sunitinib + Erlotinib (Amended Lead-In Arm B)
Number analyzed (Participants) | 8
Hours
  Cycle 1, Day 1 | 6.00 [4.00 to 8.00]
  Cycle 1, Day 15 | 5.00 [4.00 to 24.00]

27. Secondary Outcome: Dose-Corrected Observed Plasma Trough Concentrations (Ctrough) for Erlotinib on Day 1 of Cycles 3-13 (Original and Amended, Arms A and B), and Day 1 of Cycles 1-18 (Randomized)
Description: Ctrough = plasma concentration of erlotinib prior to study drug administration. Dose correction was made to the initial intended dose in Cycle 1. Assessed in the Original and Amended Lead-In (Arms A and B) Cohorts predose on Day 1 (Cycles 3-13) and in the Randomized Cohort (Sunitinib + Erlotinib treatment group only) predose on Day 1 of Cycles 1-18.
Time Frame: predose Day 1 (Cycles 3-13); predose Day 1 (Cycles 1-18)
Population: Number of participants analyzed (N)=participants with observations above lower limit of quantification (LLOQ) in Original Lead-In Cohort, Amended Lead-In Cohort (Arms A and B), Randomized Cohort (Sunitinib + Erlotinib treatment group only); n=number of participants with observations above LLOQ for specified cycle
Measure: Mean (Standard Deviation); unit: mcg/mL
Groups:
- Sunitinib + Erlotinib (All Combined): Combined Data from all participants in the Original Lead-In Cohort, Amended Lead-In Cohort (Arms A and B), and Randomized Cohort
Arm/Group | Sunitinib + Erlotinib (All Combined)
Number analyzed (Participants) | 45
mcg/mL
  Cycle 2, Day 1 (n=45) | 1.46 (0.90)
  Cycle 3, Day 1 (n=44) | 1.07 (0.76)
  Cycle 4, Day 1 (n=31) | 1.11 (0.85)
  Cycle 5, Day 1 (n=22) | 1.00 (0.93)
  Cycle 6, Day 1 (n=18) | 1.00 (0.80)
  Cycle 7, Day 1 (n=15) | 1.16 (1.30)
  Cycle 8, Day 1 (n=8) | 0.57 (0.34)
  Cycle 9, Day 1 (n=10) | 0.90 (0.68)
  Cycle 10, Day 1 (n=6) | 1.52 (1.48)
  Cycle 11, Day 1 (n=6) | 1.94 (3.67)
  Cycle 12, Day 1 (n=5) | 1.21 (1.18)
  Cycle 13, Day 1 (n=3) | 0.75 (0.43)

28. Secondary Outcome: Dose-Corrected Ctrough for Erlotinib on Day 15 Cycle 1 (Original), Day 1 of Cycle 3 (Original and Amended, Arms A and B), and Day 1 of Cycles 1-18 (Randomized)
Description: Ctrough = plasma concentration of erlotinib prior to study drug administration. Dose correction was made to the initial intended dose in Cycle 1. Assessed in the Original Cohort predose on Day 15 (Cycle 1, Time Zero) and Day 1 (Cycle 3), in the Amended Lead-In Cohort (Arms A and B) predose on Day 1 (Cycle 3) and in the Randomized Cohort (Sunitinib + Erlotinib treatment group only) predose on Day 1 of Cycles 1-18.
Time Frame: predose Day 15 (Cycle1); predose Day 1 (Cycle 3); predose Day 1 (Cycles 1-18)
Population: Number of participants analyzed (N)=participants with observations above LLOQ in Original Lead-In Cohort, Amended Lead-In Cohort (Arms A and B), Randomized Cohort (Sunitinib + Erlotinib treatment group only); n=number of participants with observations above LLOQ for specified cycle
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Sunitinib + Erlotinib (All Combined)
Number analyzed (Participants) | 45
mcg/mL
  Cycle 1, Day 15 (n=6) | 1.14 (0.92)
  Cycle 2, Day 1 (n=45) | 1.46 (0.90)
  Cycle 3, Day 1 (n=44) | 1.07 (0.76)
  Cycle 4, Day 1 (n=20) | 0.99 (0.71)
  Cycle 5, Day 1 (n=16) | 0.98 (0.99)
  Cycle 6, Day 1 (n=12) | 1.09 (0.85)
  Cycle 7, Day 1 (n=8) | 1.08 (1.13)
  Cycle 8, Day 1 (n=3) | 0.80 (0.36)
  Cycle 9, Day 1 (n=6) | 0.94 (0.80)
  Cycle 10, Day 1 (n=4) | 1.71 (1.73)
  Cycle 11, Day 1 (n=3) | 0.53 (0.57)
  Cycle 12, Day 1 (n=4) | 1.31 (1.34)
  Cycle 13, Day 1 (n=3) | 0.75 (0.43)

29. Secondary Outcome: Dose-Corrected Ctrough for Sunitinib on Day 1 of Cycles 3-13 (Original and Amended, Arms A and B), and Day 1 of Cycles 1-18 (Randomized)
Description: Ctrough = plasma concentration of sunitinib prior to study drug administration. Dose correction was made to the initial intended dose in Cycle 1. Assessed in the Original and Amended Lead-In (Arms A and B) Cohorts predose on Day 1 (Cycles 3-13) and in the Randomized Cohort (Sunitinib + Erlotinib treatment group only) predose on Day 1 of Cycles 1-18.
Time Frame: predose Day 1 (Cycles 3-13); predose Day 1 (Cycles 1-18)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib + Erlotinib (All Combined)
Number analyzed (Participants) | 44
ng/mL
  Cycle 2, Day 1 (n=44) | 22.94 (11.34)
  Cycle 3, Day 1 (n=43) | 21.48 (9.62)
  Cycle 4, Day 1 (n=28) | 19.93 (12.74)
  Cycle 5, Day 1 (n=22) | 18.58 (10.47)
  Cycle 6, Day 1 (n=19) | 22.07 (13.32)
  Cycle 7, Day 1 (n=15) | 24.85 (12.12)
  Cycle 8, Day 1 (n=8) | 18.44 (7.35)
  Cycle 9, Day 1 (n=9) | 14.81 (7.56)
  Cycle 10, Day 1 (n=6) | 17.17 (6.10)
  Cycle 11, Day 1 (n=6) | 21.42 (19.10)
  Cycle 12, Day 1 (n=4) | 11.67 (4.57)
  Cycle 13, Day 1 (n=3) | 19.79 (13.47)

30. Secondary Outcome: Dose-Corrected Ctrough for Sunitinib on Day 15 Cycle 1 (Original), Day 1 of Cycle 3 (Original and Amended, Arms A and B), and Day 1 of Cycles 1-18 (Randomized)
Description: Ctrough = plasma concentration of sunitinib prior to study drug administration. Dose correction was made to the initial intended dose in Cycle 1. Assessed in the Original Cohort predose on Day 15 (Cycle 1, Time Zero) and Day 1 (Cycle 3), in the Amended Lead-In Cohort (Arms A and B) predose on Day 1 (Cycle 3) and in the Randomized Cohort (Sunitinib + Erlotinib treatment group only) predose on Day 1 of Cycles 1-18.
Time Frame: predose Day 15 (Cycle 1) and Day 1 (Cycle 3); predose Day 1 (Cycle 3); predose Day 1 (Cycles 1-18)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib + Erlotinib (All Combined)
Number analyzed (Participants) | 44
ng/mL
  Cycle 1, Day 15 (n=7) | 18.80 (4.27)
  Cycle 2, Day 1 (n=44) | 22.94 (11.34)
  Cycle 3, Day 1 (n=43) | 21.48 (9.62)
  Cycle 4, Day 1 (n=19) | 20.58 (13.96)
  Cycle 5, Day 1 (n=16) | 17.26 (9.79)
  Cycle 6, Day 1 (n=13) | 20.16 (8.78)
  Cycle 7, Day 1 (n=8) | 21.97 (10.21)
  Cycle 8, Day 1 (n=4) | 13.56 (6.31)
  Cycle 9, Day 1 (n=6) | 15.17 (7.71)
  Cycle 10, Day 1 (n=4) | 15.61 (6.45)
  Cycle 11, Day 1 (n=3) | 15.24 (6.65)
  Cycle 12, Day 1 (n=3) | 11.99 (5.54)
  Cycle 13, Day 1 (n=3) | 19.79 (13.47)

31. Secondary Outcome: Dose-Corrected Ctrough for SU-012662 (Metabolite of Sunitinib) on Day 1 of Cycles 3-13 (Original and Amended, Arms A and B), and Day 1 of Cycles 1-18 (Randomized)
Description: Ctrough = plasma concentration of SU-012662 prior to study drug administration. Dose correction was made to the initial intended dose in Cycle 1. Assessed in the Original and Amended Lead-In (Arms A and B) Cohorts predose on Day 1 (Cycles 3-13) and in the Randomized Cohort (Sunitinib + Erlotinib treatment group only) predose on Day 1 of Cycles 1-18.
Time Frame: predose Day 1 (Cycles 3-13); predose Day 1 (Cycles 1-18)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib + Erlotinib (All Combined)
Number analyzed (Participants) | 44
ng/mL
  Cycle 2, Day 1 (n=44) | 21.02 (8.75)
  Cycle 3, Day 1 (n=43) | 19.26 (11.67)
  Cycle 4, Day 1 (n=28) | 15.74 (7.88)
  Cycle 5, Day 1 (n=22) | 15.38 (6.05)
  Cycle 6, Day 1 (n=19) | 15.04 (6.18)
  Cycle 7, Day 1 (n=15) | 17.13 (9.34)
  Cycle 8, Day 1 (n=8) | 12.50 (3.76)
  Cycle 9, Day 1 (n=9) | 12.24 (5.19)
  Cycle 10, Day 1 (n=6) | 14.29 (8.84)
  Cycle 11, Day 1 (n=6) | 19.35 (21.60)
  Cycle 12, Day 1 (n=4) | 11.58 (1.82)
  Cycle 13, Day 1 (n=3) | 15.60 (9.96)

32. Secondary Outcome: Dose-Corrected Ctrough for SU-012662 (Metabolite of Sunitinib) on Day 15 Cycle 1 (Original), Day 1 of Cycle 3 (Original and Amended, Arms A and B), and Day 1 of Cycles 1-18 (Randomized)
Description: Ctrough = plasma concentration of SU-012662 prior to study drug administration. Dose correction was made to the initial intended dose in Cycle 1. Assessed in the Original Cohort predose on Day 15 (Cycle 1, Time Zero) and Day 1 (Cycle 3), in the Amended Lead-In Cohort (Arms A and B) predose on Day 1 (Cycle 3) and in the Randomized Cohort (Sunitinib + Erlotinib treatment group only) predose on Day 1 of Cycles 1-18.
Time Frame: predose Day 15 (Cycle 1) and Day 1 (Cycle 3); predose Day 1 (Cycle 3); predose Day 1 (Cycles 1-18)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib + Erlotinib (All Combined)
Number analyzed (Participants) | 44
ng/mL
  Cycle 1, Day 15 (n=7) | 18.08 (6.14)
  Cycle 2, Day 1 (n=44) | 21.02 (8.75)
  Cycle 3, Day 1 (n=43) | 19.26 (11.67)
  Cycle 4, Day 1 (n=19) | 16.41 (7.74)
  Cycle 5, Day 1 (n=16) | 15.26 (4.97)
  Cycle 6, Day 1 (n=13) | 15.05 (4.95)
  Cycle 7, Day 1 (n=8) | 15.99 (5.03)
  Cycle 8, Day 1 (n=4) | 12.80 (3.94)
  Cycle 9, Day 1 (n=6) | 14.00 (5.59)
  Cycle 10, Day 1 (n=4) | 16.44 (10.57)
  Cycle 11, Day 1 (n=3) | 11.98 (3.31)
  Cycle 12, Day 1 (n=3) | 11.26 (2.08)
  Cycle 13, Day 1 (n=3) | 15.60 (9.96)

33. Secondary Outcome: Percentage of Participants With Epidermal Growth Factor Receptor (EGFR) Expression by Immunohistochemistry (IHC) Using 0 Percent [%] Cutoff
Description: Percentage of participants with EGFR expression by IHC using a 0% cutoff; Reported as positive, negative, or unmeasured (where positive was greater than 0% of cells demonstrating membranous staining for EGFR). Correlative analysis of EGFR expression was conducted using tumor biopsy samples collected at the time of initial diagnosis (preferred) or at the time of most recent recurrence/progression, although any time was acceptable.
Time Frame: Baseline
Population: FA Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Percentage of Participants
  Positive | 35 | 36
  Negative | 38 | 36
  Unmeasured | 26 | 28

34. Secondary Outcome: PFS in Subgroups That Were Defined by EGFR Expression (Using 0% Cutoff)
Description: PFS defined as time in weeks from date of randomization to date of first documentation of PD or death on-study due to any cause, whichever occurred first, in the following subgroups: positive, negative, or unmeasured EGFR expression. EGFR expression was analyzed using a 0% cutoff where positive was greater than 0% of cells demonstrating membranous staining for EGFR. PFS calculated as (first event date minus randomization date plus 1) divided by 7.02.
Time Frame: From randomization to Weeks 8 and 12, then every 8 weeks until disease progression or death (up to Month 17)
Population: FA Set
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Weeks
  Positive | 16.0 [7.80 to NA] — upper limit of 95 percent confidence interval was not calculable due to the large number of censored event times | 11.7 [7.10 to 13.00]
  Negative | 8.1 [7.40 to 19.10] | 8.5 [7.80 to 19.20]
  Unmeasured | 12.3 [7.70 to 43.90] | 8.4 [8.00 to 20.40]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Positive EGFR Expression; Test type: Superiority or Other; p = 0.2247, Log Rank; Hazard Ratio, log = 0.748, 95% CI 2-sided [0.351 to 1.591]
Statistical Analysis 2: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Negative EGFR Expression; Test type: Superiority or Other; p = 0.6797, Log Rank; Hazard Ratio (HR) = 1.184, 95% CI 2-sided [0.581 to 2.414]
Statistical Analysis 3: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Unmeasured EGFR Expression; Test type: Superiority or Other; p = 0.1693, Log Rank; Hazard Ratio (HR) = 0.632, 95% CI 2-sided [0.245 to 1.627]

35. Secondary Outcome: Percentage of Participants With EGFR Expression by IHC (Using 10% Cutoff)
Description: Percentage of participants with EGFR Expression by IHC using a 10% cutoff; Reported as positive (positive values were defined as being greater than 10% of cells demonstrating membranous staining for EGFR), negative, or unmeasured. Correlative analysis of EGFR expression was conducted using tumor biopsy samples collected at the time of initial diagnosis (preferred) or at the time of most recent recurrence/progression, although any time was acceptable.
Time Frame: Baseline
Population: FA Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Percentage of Participants
  Positive | 45 | 54
  Negative | 29 | 18
  Unmeasured | 26 | 28

36. Secondary Outcome: PFS in Subgroups That Were Defined by EGFR Expression (Using 10% Cutoff)
Description: PFS defined as time in weeks from date of randomization to date of first documentation of PD or death on-study due to any cause, whichever occurred first, in the following subgroups: positive, negative, or unmeasured EGFR expression. EGFR expression was analyzed using a 10% cutoff where positive was greater than 10% of cells demonstrating membranous staining for EGFR. PFS calculated as (first event date minus randomization date plus 1) divided by 7.02.
Time Frame: From randomization to Weeks 8 and 12, then every 8 weeks until disease progression or death (up to Month 17)
Population: FA Set
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Weeks
  Positive | 16.0 [7.80 to 19.50] | 10.4 [7.70 to 13.00]
  Negative | 8.1 [5.40 to 20.10] | 8.1 [4.00 to 10.10]
  Unmeasured | 12.3 [7.70 to 43.90] | 8.4 [8.00 to 20.40]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Positive EGFR Expression; Test type: Superiority or Other; p = 0.3223, Log Rank; Hazard Ratio (HR) = 0.864, 95% CI 2-sided [0.458 to 1.628]
Statistical Analysis 2: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Negative EGFR Expression; Test type: Superiority or Other; p = 0.4608, Log Rank; Hazard Ratio (HR) = 0.946, 95% CI 2-sided [0.362 to 2.474]
Statistical Analysis 3: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Unmeasured EGFR Expression; Test type: Superiority or Other; p = 0.1693, Log Rank; Hazard Ratio (HR) = 0.632, 95% CI 2-sided [0.245 to 1.627]

37. Secondary Outcome: Percentage of Participants With EGFR Gene Copy Number Increase
Description: The number of copies corresponding to exon 19 of the EGFR gene was determined by real-time quantitative polymerase chain reaction (PCR). The percentage of participants with EGFR Gene Copy Number Increase (defined as greater than 4 copies) was determined using deoxyribonucleic acid (DNA) from tumor biopsy samples collected at the time of initial diagnosis (preferred) or at the time of most recent recurrence/progression, although any time was acceptable. Reported as yes, no or unmeasured.
Time Frame: Baseline
Population: FA Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Percentage of Participants
  Yes | 0 | 1
  No | 48 | 42
  Unmeasured | 52 | 57

38. Secondary Outcome: PFS in Subgroups That Were Defined by EGFR Gene Copy Number Increase
Description: PFS, defined as time from date of randomization to the date of the first documentation of PD or death on-study due to any cause, whichever occurred first, in subgroups that were defined by EGFR gene copy number increase (reported as yes, no, or unmeasured). The number of copies corresponding to exon 19 of the EGFR gene was determined and an increase was defined as greater than 4 copies. PFS was calculated as (first event date minus randomization date plus 1)/7.02.
Time Frame: From randomization to Weeks 8 and 12, then every 8 weeks until disease progression or death (up to Month 17)
Population: FA Set
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Weeks
  Yes | NA [NA to NA] — Number of participants in category was 0 | NA [NA to NA] — Number of participants in category was 0
  No | 12.3 [8.10 to 19.10] | 8.8 [7.80 to 19.50]
  Unmeasured | 12.0 [7.70 to 43.90] | 8.1 [7.70 to 12.30]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; No EGFR Gene Copy Number Increase; Test type: Superiority or Other; p = 0.5526, Log Rank; Hazard Ratio (HR) = 1.049, 95% CI 2-sided [0.542 to 2.031]
Statistical Analysis 2: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Unmeasured EGFR Gene Copy Number Increase; Test type: Superiority or Other; p = 0.1529, Log Rank; Hazard Ratio (HR) = 0.715, 95% CI 2-sided [0.380 to 1.344]

39. Secondary Outcome: Percentage of Participants With EGFR Gene Amplification
Description: The percentage of participants with EGFR gene amplification (defined as greater than 15) was determined and reported as yes, no, or unmeasured. Correlative analysis of EGFR gene amplification was conducted using tumor biopsy samples collected at the time of initial diagnosis (preferred) or at the time of most recent recurrence/progression, although any time was acceptable.
Time Frame: Baseline
Population: FA Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Percentage of Participants
  Yes | 0 | 0
  No | 48 | 43
  Unmeasured | 52 | 57

40. Secondary Outcome: PFS in Subgroups That Were Defined by EGFR Gene Amplification
Description: PFS, defined as time from date of randomization to date of first documentation of PD or death on-study due to any cause, whichever occurred first, in subgroups that were defined by EGFR gene amplification (defined as greater than 15) and reported as no or unmeasured. PFS was calculated as (first event date minus randomization date plus 1) divided by 7.02.
Time Frame: From randomization to Weeks 8 and 12, then every 8 weeks until disease progression or death (up to Month 17)
Population: FA Set
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Weeks
  No | 12.3 [8.10 to 19.10] | 11.7 [7.80 to 52.00]
  Unmeasured | 12.0 [7.70 to 43.90] | 8.1 [7.70 to 12.30]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; No EGFR Gene Amplification; Test type: Superiority or Other; p = 0.5839, Log Rank; Hazard Ratio (HR) = 1.078, 95% CI 2-sided [0.557 to 2.085]
Statistical Analysis 2: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Unmeasured EGFR Gene Amplification; Test type: Superiority or Other; p = 0.1529, Log Rank; Hazard Ratio (HR) = 0.715, 95% CI 2-sided [0.380 to 1.344]

41. Secondary Outcome: Percentage of Participants With EGFR Gene Mutation
Description: Mutations in exons 18 through 21 of the EGFR gene were analyzed by high-performance liquid chromatography using DNA from tumor biopsy samples collected at the time of initial diagnosis (preferred) or at the time of most recent recurrence/progression, although any time was acceptable. The percentage of participants with EGFR mutations categorized as mutated, wild type or indeterminate was reported.
Time Frame: Baseline
Population: FA Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Percentage of Participants
  Mutated | 6 | 1
  Wild Type | 32 | 28
  Indeterminate | 62 | 70

42. Secondary Outcome: PFS in Subgroups That Were Defined by EGFR Gene Mutation
Description: PFS, defined as time from date of randomization to date of first documentation of PD or to death on-study due to any cause, whichever occurred first, in subgroups that were defined by EGFR gene mutation (reported as mutated, wild type, or indeterminate). PFS was calculated as (first event date minus randomization date plus 1) divided by 7.02.
Time Frame: From randomization to Weeks 8 and 12, then every 8 weeks until disease progression or death (up to Month 17)
Population: FA Set
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Weeks
  Mutated | 19.1 [3.60 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times | NA [NA to NA] — data were not calculable as only 1 participant had an event
  Wild Type | 9.0 [7.80 to 19.50] | 11.7 [4.80 to 19.50]
  Indeterminate | 12.0 [7.80 to 20.70] | 8.1 [7.70 to 12.30]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Wild Type EGFR Gene Mutation; Test type: Superiority or Other; p = 0.6324, Log Rank; Hazard Ratio (HR) = 1.160, 95% CI 2-sided [0.516 to 2.608]
Statistical Analysis 2: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Indeterminate EGFR Gene Mutation; Test type: Superiority or Other; p = 0.2413, Log Rank; Hazard Ratio (HR) = 0.813, 95% CI 2-sided [0.464 to 1.424]

43. Secondary Outcome: Percentage of Participants With KRAS (V-Ki-ras2 Kirsten Rat Sarcoma Viral Oncogene Homolog) Gene Mutations
Description: Mutations in exons 2-3 of the KRAS gene (including codons 12, 13, and 61) were analyzed by high-performance liquid chromatography using DNA from tumor biopsy samples collected at the time of initial diagnosis (preferred) or at the time of most recent recurrence/progression, although any time was acceptable. The percentage of participants with KRAS mutations categorized as mutated, wild type or indeterminate was reported.
Time Frame: Baseline
Population: FA Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Percentage of Participants
  Mutated | 9 | 6
  Wild Type | 34 | 28
  Indeterminate | 57 | 66

44. Secondary Outcome: PFS in Subgroups That Were Defined by KRAS Gene Mutation
Description: PFS, defined as time from date of randomization to date of first documentation of PD or death on-study due to any cause, whichever occurred first, in subgroups that were defined by KRAS gene mutation (reported as mutated, wild type, or indeterminate). PFS was calculated as (first event date minus randomization date plus 1) divided by 7.02.
Time Frame: From randomization to Weeks 8 and 12, then every 8 weeks until disease progression or death (up to Month 17)
Population: FA Set
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Weeks
  Mutated | 20.1 [1.40 to 20.10] | 7.5 [4.80 to 8.40]
  Wild Type | 9.5 [7.80 to 19.10] | 12.1 [7.80 to 52.00]
  Indeterminate | 12.3 [7.80 to 43.90] | 8.3 [8.00 to 12.80]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Mutated KRAS Gene Mutation; Test type: Superiority or Other; p = 0.2077, Log Rank; Hazard Ratio (HR) = 0.481, 95% CI 2-sided [0.079 to 2.910]
Statistical Analysis 2: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Wild Type KRAS Gene Mutation; Test type: Superiority or Other; p = 0.6439, Log Rank; Hazard Ratio (HR) = 1.162, 95% CI 2-sided [0.534 to 2.531]
Statistical Analysis 3: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Indeterminate KRAS Gene Mutation; Test type: Superiority or Other; p = 0.2664, Log Rank; Hazard Ratio (HR) = 0.825, 95% CI 2-sided [0.457 to 1.489]

45. Secondary Outcome: Percentage of Participants With Germline Vascular Endothelial Growth Factor Receptor 2 (VEGFR2) Polymorphisms
Description: Blood samples were collected at baseline for multiplex reverse transcription (RT) analysis of genes expressing proteins that are targets of sunitinib or involved in angiogenesis or tumor growth to determine expression levels. Percentage of participants with germline VEGFR2 single nucleotide polymorphisms (SNPs) was reported for the following genotype frequencies: homozygous C alleles (C/C), T alleles (T/T), G alleles (G/G), or A alleles (A/A), and the following heterozygous genotypes C/T, G/T, T/A, and G/A.
Time Frame: Baseline
Population: Full Analysis - All Population: all participants from lead-in period and Phase 2 (randomized phase)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- All Participants: All participants in all phases.
Arm/Group | All Participants
Number analyzed (Participants) | 162
Percentage of Participants
  Locus: VEGFR2 / rs1531289; Genotype: C/C | 44.9 [36.3 to 53.6]
  Locus: VEGFR2 / rs1531289; Genotype: C/T | 45.6 [37.0 to 54.3]
  Locus: VEGFR2 / rs1531289; Genotype: T/T | 9.6 [5.2 to 15.8]
  Locus: VEGFR2 / rs2305945; Genotype: G/G | 44.1 [35.6 to 52.9]
  Locus: VEGFR2 / rs2305945; Genotype: G/T | 47.1 [38.4 to 55.8]
  Locus: VEGFR2 / rs2305945; Genotype: T/T | 8.8 [4.6 to 14.9]
  Locus VEGFR2 / rs1870377; Genotype: T/T | 53.7 [44.9 to 62.3]
  Locus VEGFR2 / rs1870377; Genotype: T/A | 39.7 [31.4 to 48.4]
  Locus VEGFR2 / rs1870377; Genotype: A/A | 6.6 [3.1 to 12.2]
  Locus: VEGFR2 / rs2305948; Genotype: C/C | 81.6 [74.1 to 87.7]
  Locus: VEGFR2 / rs2305948; Genotype: C/T | 17.6 [11.6 to 25.1]
  Locus: VEGFR2 / rs2305948; Genotype: T/T | 0.7 [0.0 to 4.0]
  Locus: VEGFR2 / rs7692791; Genotype: C/C | 19.9 [13.5 to 27.6]
  Locus: VEGFR2 / rs7692791; Genotype: C/T | 50.7 [42.0 to 59.4]
  Locus: VEGFR2 / rs7692791; Genotype: T/T | 29.4 [21.9 to 37.8]
  Locus: VEGFR2 / rs35636987; Genotype: C/C | 100 [97.3 to 100]
  Locus: VEGFR2 / rs7667298; Genotype: C/C | 27.2 [19.9 to 35.5]
  Locus: VEGFR2 / rs7667298; Genotype: C/T | 50.0 [41.3 to 58.7]
  Locus: VEGFR2 / rs7667298; Genotype: T/T | 22.8 [16.0 to 30.8]
  Locus: VEGFR2 / rs41408948; Genotype: G/A | 57.4 [48.6 to 65.8]
  Locus: VEGFR2 / rs41408948; Genotype: A/A | 36.0 [28.0 to 44.7]
  Locus: VEGFR2 / rs41408948; Genotype: G/G | 6.6 [3.1 to 12.2]
  Locus: VEGFR2 / rs2071559; Genotype: G/G | 26.5 [19.3 to 34.7]
  Locus: VEGFR2 / rs2071559; Genotype: G/A | 47.8 [39.2 to 56.5]
  Locus: VEGFR2 / rs2071559; Genotype: A/A | 25.7 [18.6 to 33.9]

46. Secondary Outcome: PFS in Subgroups That Were Defined by Germline VEGFR2 Polymorphisms
Description: PFS, defined as time from date of randomization to date of first documentation of PD or death on-study due to any cause, whichever occurred first, in subgroups that were defined by VEGFR2 polymorphisms. PFS was calculated as (first event date minus randomization date plus 1) divided by 7.02.
Time Frame: From randomization to Weeks 8 and 12, then every 8 weeks until disease progression or death (up to Month 17)
Population: Per Protocol Caucasian Population: all Caucasian participants in randomized phase who received at least 1 dose of study medication (either erlotinib or blinded medication), with treatment assignments designated according to actual study medication received
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- Sunitinib + Erlotinib: Erlotinib 150 mg oral tablets QD in a continuous regimen expressed in 4-week cycles and Sunitinib 37.5 mg oral capsules QD in a continuous regimen expressed in 4-week cycles.
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 53 | 50
Weeks
  Locus: VEGFR2/rs1531289 Genotype: C/C | 9.00 [4.70 to 20.50] | 8.10 [7.70 to 12.80]
  Locus: VEGFR2/rs1531289 Genotype: C/T | 17.00 [7.80 to 20.10] | 8.00 [4.80 to 19.20]
  Locus: VEGFR2/rs1531289 Genotype: T/T | NA [5.40 to NA] — Values were not calculable due to the large number of censored event times | 13.00 [4.70 to NA] — Upper limit of the confidence interval was not calculable due to the large number of censored event times
  Locus: VEGFR2/rs2305945 Genotype: G/G | 17.00 [7.80 to 20.10] | 12.30 [7.50 to 13.00]
  Locus: VEGFR2/rs2305945 Genotype: G/T | 9.00 [5.30 to NA] — Upper limit of the confidence interval was not calculable due to the large number of censored event times | 7.80 [7.10 to 11.70]
  Locus: VEGFR2/rs2305945 Genotype: T/T | 20.50 [8.10 to 43.90] | NA [NA to NA] — Number of participants with an event in this category was 0
  Locus: VEGFR2/rs1870377 Genotype: T/T | 8.10 [7.80 to 20.50] | 8.00 [7.10 to 19.20]
  Locus: VEGFR2/rs1870377 Genotype: T/A | 17.00 [9.50 to 19.50] | 8.00 [5.00 to 12.10]
  Locus: VEGFR2/rs1870377 Genotype: A/A | NA [7.70 to NA] — Values were not calculable due to the large number of censored event times | 20.40 [7.50 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times
  Locus: VEGFR2/rs2305948 Genotype: C/C | 12.00 [8.10 to 20.10] | 8.00 [7.50 to 12.80]
  Locus: VEGFR2/rs2305948 Genotype: C/T | 12.30 [4.70 to 20.70] | 8.00 [7.80 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times
  Locus: VEGFR2/rs2305948 Genotype: T/T | NA [NA to NA] — Number of participants with an event in this category was 0 | 12.10 [NA to NA] — Number of participants with an event in this category was 1
  Locus: VEGFR2/rs7692791 Genotype: C/C | 12.00 [8.10 to 20.10] | 7.70 [4.70 to 19.20]
  Locus: VEGFR2/rs7692791 Genotype: C/T | 9.00 [7.80 to 43.90] | 8.50 [8.00 to 20.40]
  Locus: VEGFR2/rs7692791 Genotype: T/T | 16.00 [4.10 to 20.50] | 7.70 [4.70 to 12.10]
  Locus: VEGFR2/rs35636987 Genotype: C/C | 12.30 [8.10 to 19.50] | 8.00 [7.70 to 12.30]
  Locus: VEGFR2/rs7667298 Genotype: C/C | 12.00 [5.40 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times | 8.05 [7.50 to 12.30]
  Locus: VEGFR2/rs7667298 Genotype: C/T | 17.00 [7.80 to 20.70] | 7.80 [5.00 to 12.30]
  Locus: VEGFR2/rs7667298 Genotype: T/T | 9.50 [7.80 to 19.10] | 12.80 [4.70 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times
  Locus: VEGFR2/rs41408948 Genotype: G/G | 12.00 [7.70 to 20.50] | 11.70 [7.70 to 13.00]
  Locus: VEGFR2/rs41408948 Genotype: G/A | 17.00 [8.10 to 43.90] | 7.75 [4.70 to 12.30]
  Locus: VEGFR2/rs41408948 Genotype: A/A | 13.45 [7.80 to 19.10] | 13.60 [4.70 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times
  Locus: VEGFR2/rs2071559 Genotype: G/G | 9.50 [7.80 to 20.50] | 12.80 [8.00 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times
  Locus: VEGFR2/rs2071559 Genotype: G/A | 17.00 [8.10 to 43.90] | 7.80 [5.00 to 13.00]
  Locus: VEGFR2/rs2071559 Genotype: A/A | 8.10 [5.40 to 12.30] | 8.00 [7.50 to 12.30]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs1531289 Genotype: C/C; Test type: Superiority or Other; p = 0.7423, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.130, 95% CI 2-sided [0.541 to 2.360]
Statistical Analysis 2: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs1531289 Genotype: C/T; Test type: Superiority or Other; p = 0.1570, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.598, 95% CI 2-sided [0.290 to 1.236]
Statistical Analysis 3: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs1531289 Genotype: T/T; Test type: Superiority or Other; p = 0.7954, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.794, 95% CI 2-sided [0.131 to 4.819]
Statistical Analysis 4: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs2305945 Genotype: G/G; Test type: Superiority or Other; p = 0.6210, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.833, 95% CI 2-sided [0.401 to 1.732]
Statistical Analysis 5: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs2305945 Genotype: G/T; Test type: Superiority or Other; p = 0.5268, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.794, 95% CI 2-sided [0.385 to 1.640]
Statistical Analysis 6: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs1870377 Genotype: T/T; Test type: Superiority or Other; p = 0.9753, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.011, 95% CI 2-sided [0.504 to 2.027]
Statistical Analysis 7: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs1870377 Genotype: T/A; Test type: Superiority or Other; p = 0.0141, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.378, 95% CI 2-sided [0.168 to 0.850]
Statistical Analysis 8: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs1870377 Genotype: A/A; Test type: Superiority or Other; p = 0.5596, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 2.236, 95% CI 2-sided [0.139 to 35.90]
Statistical Analysis 9: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs2305948 Genotype: C/C; Test type: Superiority or Other; p = 0.2788, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.738, 95% CI 2-sided [0.422 to 1.288]
Statistical Analysis 10: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs2305948 Genotype: C/T; Test type: Superiority or Other; p = 0.8971, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.075, 95% CI 2-sided [0.352 to 3.286]
Statistical Analysis 11: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs7692791 Genotype: C/C; Test type: Superiority or Other; p = 0.6559, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.775, 95% CI 2-sided [0.251 to 2.388]
Statistical Analysis 12: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs7692791 Genotype: C/T; Test type: Superiority or Other; p = 0.8563, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.939, 95% CI 2-sided [0.466 to 1.889]
Statistical Analysis 13: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs7692791 Genotype: T/T; Test type: Superiority or Other; p = 0.668, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.382, 95% CI 2-sided [0.130 to 1.120]
Statistical Analysis 14: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs35636987 Genotype: C/C; Test type: Superiority or Other; p = 0.3681, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.800, 95% CI 2-sided [0.488 to 1.309]
Statistical Analysis 15: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs7667298 Genotype: C/C; Test type: Superiority or Other; p = 0.7520, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.860, 95% CI 2-sided [0.331 to 2.237]
Statistical Analysis 16: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs7667298 Genotype: C/T; Test type: Superiority or Other; p = 0.0833, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.551, 95% CI 2-sided [0.276 to 1.098]
Statistical Analysis 17: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs7667298 Genotype: T/T; Test type: Superiority or Other; p = 0.4772, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.564, 95% CI 2-sided [0.444 to 5.506]
Statistical Analysis 18: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs41408948 Genotype: G/G; Test type: Superiority or Other; p = 0.9235, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.034, 95% CI 2-sided [0.522 to 2.048]
Statistical Analysis 19: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs41408948 Genotype: G/A; Test type: Superiority or Other; p = 0.0845, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.501, 95% CI 2-sided [0.223 to 1.126]
Statistical Analysis 20: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs41408948 Genotype: A/A; Test type: Superiority or Other; p = 0.5493, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.724, 95% CI 2-sided [0.284 to 10.47]
Statistical Analysis 21: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs2071559 Genotype: G/G; Test type: Superiority or Other; p = 0.5210, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.400, 95% CI 2-sided [0.492 to 3.987]
Statistical Analysis 22: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs2071559 Genotype: G/A; Test type: Superiority or Other; p = 0.0854, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.538, 95% CI 2-sided [0.261 to 1.108]
Statistical Analysis 23: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs2071559 Genotype: A/A; Test type: Superiority or Other; p = 0.9198, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.953, 95% CI 2-sided [0.365 to 2.489]

47. Secondary Outcome: Overall Survival (OS) in Subgroups That Were Defined by Germline VEGFR2 Polymorphisms
Description: OS, defined as time from date of randomization to date of death due to any cause, in subgroups that were defined by VEGFR2 polymorphisms. OS was calculated as (date of death minus date of randomization plus 1) divided by 30.4.
Time Frame: From randomization until death (up to Month 17)
Population: Per Protocol Caucasian Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 53 | 50
Months
  Locus: VEGFR2/rs1531289 Genotype: C/C | 8.20 [5.40 to 12.80] | 6.20 [4.40 to 14.40]
  Locus: VEGFR2/rs1531289 Genotype: C/T | 6.40 [5.20 to 11.30] | 5.30 [4.30 to 16.70]
  Locus: VEGFR2/rs1531289 Genotype: T/T | 11.60 [3.70 to 16.30] | 16.50 [1.30 to 28.80]
  Locus: VEGFR2/rs2305945 Genotype: G/G | 8.00 [5.70 to 11.30] | 5.50 [4.20 to 16.70]
  Locus: VEGFR2/rs2305945 Genotype: G/T | 6.25 [4.70 to 9.70] | 7.60 [5.30 to 13.40]
  Locus: VEGFR2/rs2305945 Genotype: T/T | NA [5.40 to NA] — Data were not calculable due to the large number of censored event times | NA [2.20 to NA] — Data were not calculable due to the large number of censored event times
  Locus: VEGFR2/rs1870377 Genotype: T/T | 6.40 [5.20 to 14.00] | 10.00 [4.90 to 17.00]
  Locus: VEGFR2/rs1870377 Genotype: T/A | 8.00 [6.30 to 11.30] | 4.70 [3.90 to 6.80]
  Locus: VEGFR2/rs1870377 Genotype: A/A | NA [4.20 to NA] — Data were not calculable due to the large number of censored event times | NA [3.90 to NA] — Data were not calculable due to the large number of censored event times
  Locus: VEGFR2/rs2305948 Genotype: C/C | 8.40 [6.20 to 12.80] | 10.00 [4.60 to 16.50]
  Locus: VEGFR2/rs2305948 Genotype: C/T | 5.80 [5.10 to 9.30] | 4.90 [4.30 to 6.80]
  Locus: VEGFR2/rs2305948 Genotype: T/T | NA [NA to NA] — Number of participants with an event (death) in this category was 0 | NA [5.90 to NA] — Data were not calculable due to the large number of censored event times
  Locus: VEGFR2/rs7692791 Genotype: C/C | 6.40 [5.40 to 11.30] | 7.60 [1.80 to 16.50]
  Locus: VEGFR2/rs7692791 Genotype: C/T | 9.30 [5.80 to 12.80] | 5.80 [4.40 to 28.80]
  Locus: VEGFR2/rs7692791 Genotype: T/T | 6.30 [4.20 to NA] — Upper limit of confidence interval was not calculable | 10.00 [4.60 to 16.70]
  Locus: VEGFR2/rs35636987 Genotype: C/C | 8.00 [5.70 to 11.30] | 6.80 [4.80 to 13.40]
  Locus: VEGFR2/rs7667298 Genotype: C/C | 9.30 [4.80 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times | 13.40 [4.60 to 16.50]
  Locus: VEGFR2/rs7667298 Genotype: C/T | 6.65 [5.20 to 9.70] | 4.90 [3.90 to 10.00]
  Locus: VEGFR2/rs7667298 Genotype: T/T | 11.30 [4.10 to 12.80] | 9.60 [4.40 to 28.80]
  Locus: VEGFR2/rs41408948 Genotype: G/G | 6.40 [5.10 to 11.60] | 8.40 [4.90 to 16.50]
  Locus: VEGFR2/rs41408948 Genotype: G/A | 8.00 [5.20 to 11.30] | 4.40 [3.90 to 16.70]
  Locus: VEGFR2/rs41408948 Genotype: A/A | 11.30 [NA to NA] — Number of participants with an event (death) equal 1 in this category | 9.55 [5.30 to 28.80]
  Locus: VEGFR2/rs2071559 Genotype: G/G | 11.30 [5.40 to 12.80] | 8.60 [4.40 to 17.00]
  Locus: VEGFR2/rs2071559 Genotype: G/A | 6.90 [5.20 to 11.30] | 4.90 [3.90 to 16.50]
  Locus: VEGFR2/rs2071559 Genotype: A/A | 9.30 [4.80 to 14.00] | 13.40 [4.60 to 14.40]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs1531289 Genotype: C/C; Test type: Superiority or Other; p = 0.9486, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.977, 95% CI 2-sided [0.473 to 2.014]
Statistical Analysis 2: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs1531289 Genotype: C/T; Test type: Superiority or Other; p = 0.9084, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.961, 95% CI 2-sided [0.487 to 1.897]
Statistical Analysis 3: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs1531289 Genotype: T/T; Test type: Superiority or Other; p = 0.2009, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 2.876, 95% CI 2-sided [0.534 to 15.48]
Statistical Analysis 4: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs2305845 Genotype: G/G; Test type: Superiority or Other; p = 0.7863, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.098, 95% CI 2-sided [0.554 to 2.175]
Statistical Analysis 5: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEFR2/rs2305945 Genotype: G/T; Test type: Superiority or Other; p = 0.5267, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.243, 95% CI 2-sided [0.633 to 2.442]
Statistical Analysis 6: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs2305945 Genotype: T/T; Test type: Superiority or Other; p = 0.6240, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.550, 95% CI 2-sided [0.049 to 6.208]
Statistical Analysis 7: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEFR/rs1870377 Genotype: T/T; Test type: Superiority or Other; p = 0.4882, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.254, 95% CI 2-sided [0.660 to 2.384]
Statistical Analysis 8: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs1870377 Genotype: T/A; Test type: Superiority or Other; p = 0.1307, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.587, 95% CI 2-sided [0.290 to 1.189]
Statistical Analysis 9: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs1870377 Genotype: A/A; Test type: Superiority or Other; p = 0.5596, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 2.236, 95% CI 2-sided [0.139 to 35.90]
Statistical Analysis 10: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs2305948 Genotype: C/C; Test type: Superiority or Other; p = 0.7966, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.073, 95% CI 2-sided [0.628 to 1.833]
Statistical Analysis 11: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs2305948 Genotype: C/T; Test type: Superiority or Other; p = 0.9224, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.954, 95% CI 2-sided [0.366 to 2.484]
Statistical Analysis 12: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs7692791 Genotype: C/C; Test type: Superiority or Other; p = 0.9317, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.047, 95% CI 2-sided [0.363 to 3.025]
Statistical Analysis 13: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs7692791 Genotype: C/T; Test type: Superiority or Other; p = 0.8696, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.057, 95% CI 2-sided [0.546 to 2.044]
Statistical Analysis 14: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs7692791 Genotype: T/T; Test type: Superiority or Other; p = 0.8694, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.075, 95% CI 2-sided [0.453 to 2.554]
Statistical Analysis 15: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs3563987 Genotype: C/C; Test type: Superiority or Other; p = 0.8708, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.039, 95% CI 2-sided [0.654 to 1.652]
Statistical Analysis 16: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs7667298 Genotype: C/C; Test type: Superiority or Other; p = 0.7667, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.157, 95% CI 2-sided [0.442 to 3.026]
Statistical Analysis 17: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs7667298 Genotype: C/T; Test type: Superiority or Other; p = 0.3822, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.755, 95% CI 2-sided [0.401 to 1.422]
Statistical Analysis 18: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs7667298 Genotype: T/T; Test type: Superiority or Other; p = 0.5089, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.419, 95% CI 2-sided [0.498 to 4.040]
Statistical Analysis 19: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs41408948 Genotype: G/G; Test type: Superiority or Other; p = 0.3944, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.326, 95% CI 2-sided [0.691 to 2.544]
Statistical Analysis 20: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs41408948 Genotype: G/A; Test type: Superiority or Other; p = 0.3103, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.692, 95% CI 2-sided [0.339 to 1.416]
Statistical Analysis 21: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs41408948 Genotype: A/A; Test type: Superiority or Other; p = 0.8942, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.857, 95% CI 2-sided [0.089 to 8.294]
Statistical Analysis 22: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs2071559 Genotype: G/G; Test type: Superiority or Other; p = 0.6650, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.240, 95% CI 2-sided [0.466 to 3.304]
Statistical Analysis 23: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs2071559 Genotype: G/A; Test type: Superiority or Other; p = 0.4415, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.779, 95% CI 2-sided [0.412 to 1.475]
Statistical Analysis 24: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: VEGFR2/rs2071559 Genotype: A/A; Test type: Superiority or Other; p = 0.4682, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.458, 95% CI 2-sided [0.523 to 4.060]

48. Secondary Outcome: Percentage of Participants With Germline Platelet-derived Growth Factor Receptor Beta (PDGFRB) Polymorphisms
Description: Blood samples were collected at baseline for multiplex RT analysis of genes expressing proteins that are targets of sunitinib or involved in angiogenesis or tumor growth to determine expression levels. Percentage of participants with germline PDGFRB SNPs was reported for the following genotype frequencies: homozygous C alleles (C/C), T alleles (T/T), G alleles (G/G), or A alleles (A/A), and the following heterozygous genotypes C/T, A/T, A/G, T/C, T/G, G/C, C/A and G/A.
Time Frame: Baseline
Population: Full Analysis - All Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | All Participants
Number analyzed (Participants) | 162
Percentage of Participants
  Locus: PDGFRB / rs2304060 Genotype:C/C | 21.3 [14.8 to 29.2]
  Locus: PDGFRB / rs2304060 Genotype: C/A | 52.9 [44.2 to 61.6]
  Locus: PDGFRB / rs2304060 Genotype: A/A | 25.7 [18.6 to 33.9]
  Locus: PDGFRB / rs17656204 Genotype: C/C | 48.5 [39.9 to 57.2]
  Locus: PDGFRB / rs17656204 Genotype: C/T | 44.1 [35.6 to 52.9]
  Locus: PDGFRB / rs17656204 Genotype: T/T | 7.4 [3.6 to 13.1]
  Locus: PDGFRB / rs2304061 Genotype: G/G | 51.9 [43.1 to 60.5]
  Locus: PDGFRB / rs2304061 Genotype: G/A | 44.4 [35.9 to 53.2]
  Locus: PDGFRB / rs2304061 Genotype: A/A | 3.7 [1.2 to 8.4]
  Locus: PDGFRB / rs1077724 Genotype: A/A | 43.4 [34.9 to 52.1]
  Locus: PDGFRB / rs1077724 Genotype: A/T | 46.3 [37.7 to 55.1]
  Locus: PDGFRB / rs1077724 Genotype: T/T | 10.3 [5.7 to 16.7]
  Locus: PDGFRB / rs919751 Genotype: A/A | 46.3 [37.7 to 55.1]
  Locus: PDGFRB / rs919751 Genotype: A/G | 39.0 [30.7 to 47.7]
  Locus: PDGFRB / rs919751 Genotype: G/G | 14.7 [9.2 to 21.8]
  Locus: PDGFRB / rs2304058 Genotype: G/G | 25.7 [18.6 to 33.9]
  Locus: PDGFRB / rs2304058 Genotype: G/C | 49.3 [40.6 to 58.0]
  Locus: PDGFRB / rs2304058 Genotype: C/C | 25.0 [18.0 to 33.1]
  Locus: PDGFRB / rs1864972 Genotype: G/G | 41.2 [32.8 to 49.9]
  Locus: PDGFRB / rs1864972 Genotype: G/A | 41.9 [33.5 to 50.7]
  Locus: PDGFRB / rs1864972 Genotype: A/A | 16.9 [11.0 to 24.3]
  Locus: PDGFRB / rs3733678 Genotype: G/G | 80.1 [72.4 to 86.5]
  Locus: PDGFRB / rs3733678 Genotype: G/A | 19.9 [13.5 to 27.6]
  Locus: PDGFRB / rs246396 Genotype: T/T | 70.6 [62.2 to 78.1]
  Locus: PDGFRB / rs246396 Genotype: T/C | 27.2 [19.9 to 35.5]
  Locus: PDGFRB / rs246396 Genotype: C/C | 2.2 [0.5 to 6.3]
  Locus: PDGFRB / rs34586048 Genotype: C/C | 100 [97.3 to 100]
  Locus: PDGFRB / rs11740355 Genotype: T/T | 80.9 [73.3 to 87.1]
  Locus: PDGFRB / rs11740355 Genotype: T/G | 18.4 [12.3 to 25.9]
  Locus: PDGFRB / rs11740355 Genotype: G/G | 0.7 [0.0 to 4.0]
  Locus: PDGFRB / rs740751 Genotype: C/C | 41.2 [32.8 to 49.9]
  Locus: PDGFRB / rs740751 Genotype: C/T | 41.2 [32.8 to 49.9]
  Locus: PDGFRB / rs740751 Genotype: T/T | 17.6 [11.6 to 25.1]
  Locus: PDGFRB / rs4705415 Genotype: G/G | 36.0 [28.0 to 44.7]
  Locus: PDGFRB / rs4705415 Genotype: G/A | 44.1 [35.6 to 52.9]
  Locus: PDGFRB / rs4705415 Genotype: A/A | 19.9 [13.5 to 27.6]
  Locus: PDGFRB / rs3776075 Genotype: T/T | 22.8 [16.0 to 30.8]
  Locus: PDGFRB / rs3776075 Genotype: T/G | 56.6 [47.9 to 65.1]
  Locus: PDGFRB / rs3776075 Genotype: G/G | 20.6 [14.1 to 28.4]
  Locus: PDGFRB / rs17708574 Genotype: G/G | 79.4 [71.6 to 85.9]
  Locus: PDGFRB / rs17708574 Genotype: G/A | 17.6 [11.6 to 25.1]
  Locus: PDGFRB / rs17708574 Genotype: A/A | 2.9 [0.8 to 7.4]
  Locus: PDGFRB / rs10063714 Genotype: T/T | 76.5 [68.4 to 83.3]
  Locus: PDGFRB / rs10063714 Genotype: T/A | 22.1 [15.4 to 30.0]
  Locus: PDGFRB / rs10063714 Genotype: A/A | 1.5 [0.2 to 5.2]
  Locus: PDGFRB / rs3776081 Genotype: A/A | 39.0 [30.7 to 47.7]
  Locus: PDGFRB / rs3776081 Genotype: A/G | 47.1 [38.4 to 55.8]
  Locus: PDGFRB / rs3776081 Genotype: G/G | 14.0 [8.6 to 21.0]
  Locus: PDGFRB / rs2007637 Genotype: G/G | 79.4 [71.6 to 85.9]
  Locus: PDGFRB / rs2007637 Genotype: G/A | 19.1 [12.9 to 26.7]
  Locus: PDGFRB / rs2007637 Genotype: A/A | 1.5 [0.2 to 5.2]
  Locus: PDGFRB / rs2302273 Genotype: G/G | 56.0 [47.1 to 64.5]
  Locus: PDGFRB / rs2302273 Genotype: G/A | 38.1 [29.8 to 46.8]
  Locus: PDGFRB / rs2302273 Genotype: A/A | 6.0 [2.6 to 11.4]

49. Secondary Outcome: PFS in Subgroups That Were Defined by Germline PDGFRB Polymorphisms
Description: PFS, defined as time from date of randomization to date of first documentation of PD or death on-study due to any cause, whichever occurred first, in subgroups that were defined by PDGFRB polymorphisms. PFS was calculated as (first event date minus randomization date plus 1) divided by 7.02.
Time Frame: From randomization to Weeks 8 and 12, then every 8 weeks until disease progression or death (up to Month 17)
Population: Per Protocol Caucasian Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 53 | 50
Weeks
  Locus: PDGFRB/rs2304060 Genotype: C/C | 12.30 [7.80 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times | 19.20 [11.7 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times
  Locus: PDGFRB/rs2304060 Genotype: C/A | 9.00 [7.70 to 20.50] | 8.00 [5.40 to 12.30]
  Locus: PDGFRB/rs2304060 Genotype: A/A | 12.00 [7.80 to 20.10] | 7.90 [7.10 to 12.80]
  Locus: PDGFRB/rs17656204 Genotype: C/C | 16.00 [7.80 to 20.50] | 8.00 [7.50 to 13.00]
  Locus: PDGFRB/rs17656204 Genotype: C/T | 17.00 [7.70 to 20.70] | 8.00 [4.80 to 11.70]
  Locus: PDGFRB/rs17656204 Genotype: T/T | 8.65 [4.00 to 12.30] | NA [NA to NA] — Number of participants with event in this category was zero
  Locus: PDGFRB/rs2304061 Genotype: G/G | 19.50 [8.10 to 20.70] | 7.80 [7.10 to 12.80]
  Locus: PDGFRB/rs2304061 Genotype: G/A | 7.80 [5.40 to 19.10] | 8.10 [7.70 to 13.00]
  Locus: PDGFRB/rs2304061 Genotype: A/A | 10.90 [9.50 to 12.30] | NA [NA to NA] — Number of participants in this category was zero
  Locus: PDGFRB/rs1077724 Genotype: A/A | 12.00 [7.80 to 20.50] | 8.00 [7.50 to 20.40]
  Locus: PDGFRB/rs1077724 Genotype: A/T | 17.00 [7.70 to 43.90] | 7.85 [4.80 to 8.50]
  Locus: PDGFRB/rs1077724 Genotype: T/T | 12.30 [9.50 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times | 19.20 [13.0 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times
  Locus: PDGFRB/rs919751 Genotype: A/A | 9.50 [5.40 to 43.90] | 11.70 [7.80 to 13.00]
  Locus: PDGFRB/rs919751 Genotype: A/G | 12.00 [7.80 to 19.10] | 7.85 [5.40 to 20.40]
  Locus: PDGFRB/rs919751 Genotype: G/G | 19.50 [7.80 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times | 7.70 [4.00 to 12.80]
  Locus: PDGFRB/rs2304058 Genotype: G/G | 19.50 [7.80 to 43.90] | 6.35 [4.00 to 12.80]
  Locus: PDGFRB/rs2304058 Genotype: G/C | 9.00 [7.80 to 20.50] | 8.00 [7.50 to 19.20]
  Locus: PDGFRB/rs2304058 Genotype: C/C | 12.30 [5.40 to 19.10] | 8.50 [8.00 to 12.10]
  Locus: PDGFRB/rs1864975 Genotype: G/G | 20.10 [7.80 to 20.70] | 7.85 [4.70 to 52.00]
  Locus: PDGFRB/rs1864975 Genotype: G/A | 8.10 [7.40 to 17.00] | 8.00 [7.50 to 13.00]
  Locus: PDGFRB/rs1864975 Genotype: A/A | 12.30 [9.50 to 19.10] | 8.10 [4.70 to 11.70]
  Locus: PDGFRB/rs3733678 Genotype: G/G | 12.00 [8.10 to 19.10] | 8.00 [7.50 to 11.70]
  Locus: PDGFRB/rs3733678 Genotype: G/A | 20.50 [5.40 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times | NA [12.1 to NA] — Data were not calculable due to the large number of censored event times
  Locus: PDGFRB/rs246396 Genotype: T/T | 16.00 [8.10 to 20.70] | 8.00 [7.10 to 12.30]
  Locus: PDGFRB/rs246396 Genotype: T/C | 7.80 [4.30 to 19.10] | 8.10 [7.50 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times
  Locus: PDGFRB/rs246396 Genotype: C/C | 12.30 [NA to NA] — Confidence interval was not calculable due to the large number of censored event times | 8.00 [NA to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times
  Locus: PDGFRB/rs34586048 Genotype: C/C | 12.30 [8.10 to 19.50] | 8.00 [7.70 to 12.30]
  Locus: PDGFRB/rs11740355 Genotype: T/T | 12.30 [7.80 to 20.50] | 8.50 [7.70 to 12.30]
  Locus: PDGFRB/rs11740355 Genotype: T/G | 16.00 [8.10 to 19.50] | 7.40 [4.70 to NA] — Upper limit of the confidence interval was not calculable due to the large number of censored event times
  Locus: PDGFRB/rs11740355 Genotype: G/G | 7.80 [NA to NA] — Number of participants in this category was 1 | NA [NA to NA] — Number of participants in this category was zero
  Locus: PDGFRB/rs740751 Genotype: C/C | 20.10 [7.80 to 20.70] | 8.00 [4.70 to 52.00]
  Locus: PDGFRB/rs740751 Genotype: C/T | 8.10 [7.40 to 17.00] | 8.00 [7.50 to 13.00]
  Locus: PDGFRB/rs740751 Genotype: T/T | 12.30 [9.50 to 19.10] | 8.10 [4.70 to 11.70]
  Locus: PDGFRB/rs4705415 Genotype: G/G | 19.10 [9.50 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times | 11.70 [8.00 to 19.20]
  Locus: PDGFRB/rs4705415 Genotype: G/A | 8.10 [7.80 to 20.50] | 7.90 [7.50 to 12.30]
  Locus: PDGFRB/rs4705415 Genotype: A/A | 19.50 [7.80 to 20.70] | 7.70 [4.00 to 12.80]
  Locus: PDGFRB/rs3776075 Genotype: T/T | 16.00 [4.10 to 20.10] | 7.50 [5.00 to 12.80]
  Locus: PDGFRB/rs3776075 Genotype: T/G | 12.00 [8.10 to 20.50] | 8.05 [7.80 to 13.00]
  Locus: PDGFRB/rs3776075 Genotype: G/G | NA [5.30 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times | 10.10 [4.70 to 19.20]
  Locus: PDGFRB/rs17708574 Genotype: G/G | 12.30 [8.10 to 20.10] | 8.05 [7.50 to 12.80]
  Locus: PDGFRB/rs17708574 Genotype: G/A | 9.00 [4.10 to 20.70] | 7.90 [7.50 to 12.30]
  Locus: PDGFRB/rs10063714 Genotype: T/T | 12.00 [8.10 to 19.10] | 8.00 [7.50 to 8.50]
  Locus: PDGFRB/rs10063714 Genotype: T/A | 20.50 [5.40 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times | 19.20 [12.1 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times
  Locus: PDGFRB/rs3776081 Genotype: A/A | 19.50 [7.80 to 20.70] | 7.70 [5.00 to 12.80]
  Locus: PDGFRB/rs3776081 Genotype: A/G | 12.00 [8.10 to 19.10] | 8.10 [7.80 to 20.40]
  Locus: PDGFRB/rs3776081 Genotype: G/G | NA [5.30 to NA] — Data were not calculable due to the large number of censored event times | 10.10 [4.70 to 12.10]
  Locus: PDGFRB/rs2007637 Genotype: G/G | 16.00 [8.10 to 20.50] | 8.00 [7.50 to 12.10]
  Locus: PDGFRB/rs2007637 Genotype: G/A | 12.30 [7.80 to 20.10] | 12.80 [7.50 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times
  Locus: PDGFRB/rs2007637 Genotype: A/A | 4.30 [NA to NA] — Number of participants in this category was 1 | 52.00 [NA to NA] — Number of participants in this category was 1
  Locus: PDGFRB/rs2302273 Genotype: G/G | 19.50 [7.80 to 20.70] | 10.15 [7.50 to 19.20]
  Locus: PDGFRB/rs2302273 Genotype: G/A | 9.50 [7.80 to 17.00] | 8.00 [7.10 to 12.30]
  Locus: PDGFRB/rs2302273 Genotype: A/A | NA [5.30 to NA] — Data were not calculable due to the large number of censored event times | 10.10 [4.70 to 12.10]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2304060 Genotype: C/C; Test type: Superiority or Other; p = 0.7301, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.289, 95% CI 2-sided [0.304 to 5.470]
Statistical Analysis 2: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; PDGFRB/rs2304060 C/A; Test type: Superiority or Other; p = 0.5013, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.788, 95% CI 2-sided [0.390 to 1.592]
Statistical Analysis 3: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2304060 Genotype: A/A; Test type: Superiority or Other; p = 0.3680, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.686, 95% CI 2-sided [0.298 to 1.578]
Statistical Analysis 4: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs17656204 Genotype: C/C; Test type: Superiority or Other; p = 0.3804, Log Rank — 2-sided, unstratified log-rank test; Hazard Ratio (HR) = 0.738, 95% CI 2-sided [0.371 to 1.467]
Statistical Analysis 5: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs17656204 Genotype: C/T; Test type: Superiority or Other; p = 0.1507, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.570, 95% CI 2-sided [0.261 to 1.247]
Statistical Analysis 6: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus PDGFRB/rs17656204 Genotype: T/T; Test type: Superiority or Other; p = 0.0772, Log Rank — 2-sided unstratified log-rank test
Statistical Analysis 7: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2304061 Genotype: G/G; Test type: Superiority or Other; p = 0.2149, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.660, 95% CI 2-sided [0.339 to 1.284]
Statistical Analysis 8: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/RS2304061 Genotype: G/A; Test type: Superiority or Other; p = 0.9491, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.026, 95% CI 2-sided [0.466 to 2.260]
Statistical Analysis 9: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs1077724 Genotype: A/A; Test type: Superiority or Other; p = 0.8114, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.917, 95% CI 2-sided [0.447 to 1.881]
Statistical Analysis 10: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs1077724 Genotype: A/T; Test type: Superiority or Other; p = 0.1379, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.577, 95% CI 2-sided [0.273 to 1.221]
Statistical Analysis 11: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs1077724 Genotype: T/T; Test type: Superiority or Other; p = 0.5341, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.859, 95% CI 2-sided [0.256 to 13.51]
Statistical Analysis 12: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs919751 Genotype: A/A; Test type: Superiority or Other; p = 0.8564, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.932, 95% CI 2-sided [0.431 to 2.014]
Statistical Analysis 13: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs919751 Genotype: A/G; Test type: Superiority or Other; p = 0.5766, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.797, 95% CI 2-sided [0.355 to 1.788]
Statistical Analysis 14: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs919751 Genotype: G/G; Test type: Superiority or Other; p = 0.2043, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.467, 95% CI 2-sided [0.140 to 1.557]
Statistical Analysis 15: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2304058 Genotype: G/G; Test type: Superiority or Other; p = 0.1626, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.531, 95% CI 2-sided [0.214 to 1.317]
Statistical Analysis 16: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2304058 Genotype: G/C; Test type: Superiority or Other; p = 0.9680, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.986, 95% CI 2-sided [0.484 to 2.006]
Statistical Analysis 17: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2304058 Genotype: C/C; Test type: Superiority or Other; p = 0.3587, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.573, 95% CI 2-sided [0.171 to 1.920]
Statistical Analysis 18: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs1864972 Genotype: G/G; Test type: Superiority or Other; p = 0.4635, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.742, 95% CI 2-sided [0.331 to 1.662]
Statistical Analysis 19: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs1864972 Genotype: G/A; Test type: Superiority or Other; p = 0.9834, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.992, 95% CI 2-sided [0.476 to 2.069]
Statistical Analysis 20: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs1864972 Genotype: A/A; Test type: Superiority or Other; p = 0.1764, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.353, 95% CI 2-sided [0.072 to 1.725]
Statistical Analysis 21: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs3733678 Genotype: G/G; Test type: Superiority or Other; p = 0.2018, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.715, 95% CI 2-sided [0.422 to 1.209]
Statistical Analysis 22: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs3733678 Genotype: G/A; Test type: Superiority or Other; p = 0.4592, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.850, 95% CI 2-sided [0.354 to 9.673]
Statistical Analysis 23: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs246396 Genotype: T/T; Test type: Superiority or Other; p = 0.1593, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.665, 95% CI 2-sided [0.373 to 1.184]
Statistical Analysis 24: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs246396 Genotype: T/C; Test type: Superiority or Other; p = 0.5897, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.327, 95% CI 2-sided [0.469 to 3.755]
Statistical Analysis 25: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs34586048 Genotype: C/C; Test type: Superiority or Other; p = 0.3681, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.800, 95% CI 2-sided [0.488 to 1.309]
Statistical Analysis 26: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs11740355 Genotype: T/T; Test type: Superiority or Other; p = 0.3235, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.752, 95% CI 2-sided [0.423 to 1.336]
Statistical Analysis 27: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs11740355 Genotype: T/G; Test type: Superiority or Other; p = 0.7463, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.845, 95% CI 2-sided [0.303 to 2.355]
Statistical Analysis 28: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: rs740751 Genotype: C/C; Test type: Superiority or Other; p = 0.4179, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.724, 95% CI 2-sided [0.330 to 1.593]
Statistical Analysis 29: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs740751 Genotype: C/T; Test type: Superiority or Other; p = 0.9423, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.973, 95% CI 2-sided [0.462 to 2.050]
Statistical Analysis 30: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs7407451 Genotype: T/T; Test type: Superiority or Other; p = 0.1764, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.353, 95% CI 2-sided [0.072 to 1.725]
Statistical Analysis 31: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs4705415 Genotype: G/G; Test type: Superiority or Other; p = 0.2352, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.549, 95% CI 2-sided [0.201 to 1.501]
Statistical Analysis 32: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs4705415 Genotype: G/A; Test type: Superiority or Other; p = 0.9674, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.986, 95% CI 2-sided [0.485 to 2.003]
Statistical Analysis 33: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs4705415 Genotype: A/A; Test type: Superiority or Other; p = 0.3524, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.629, 95% CI 2-sided [0.235 to 1.686]
Statistical Analysis 34: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs3776075 Genotype: T/T; Test type: Superiority or Other; p = 0.6652, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.809, 95% CI 2-sided [0.308 to 2.124]
Statistical Analysis 35: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs3776075 Genotype: T/G; Test type: Superiority or Other; p = 0.5931, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.839, 95% CI 2-sided [0.436 to 1.618]
Statistical Analysis 36: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs3776075 Genotype: G/G; Test type: Superiority or Other; p = 0.2625, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.475, 95% CI 2-sided [0.125 to 1.813]
Statistical Analysis 37: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs17708574 Genotype: G/G; Test type: Superiority or Other; p = 0.2168, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.704, 95% CI 2-sided [0.400 to 1.239]
Statistical Analysis 38: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs17708574 Genotype: G/A; Test type: Superiority or Other; p = 0.9802, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.987, 95% CI 2-sided [0.353 to 2.759]
Statistical Analysis 39: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs10063714 Genotype: T/T; Test type: Superiority or Other; p = 0.1145, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.652, 95% CI 2-sided [0.378 to 1.122]
Statistical Analysis 40: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs10063714 Genotype: T/A; Test type: Superiority or Other; p = 0.7725, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.192, 95% CI 2-sided [0.360 to 3.946]
Statistical Analysis 41: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs3776081 Genotype: A/A; Test type: Superiority or Other; p = 0.3286, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.687, 95% CI 2-sided [0.321 to 1.473]
Statistical Analysis 42: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs3776081 Genotype: A/G; Test type: Superiority or Other; p = 0.9480, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.976, 95% CI 2-sided [0.470 to 2.028]
Statistical Analysis 43: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs3776081 Genotype: G/G; Test type: Superiority or Other; p = 0.3844, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.531, 95% CI 2-sided [0.125 to 2.282]
Statistical Analysis 44: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2007637 Genotype: G/G; Test type: Superiority or Other; p = 0.1373, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.662, 95% CI 2-sided [0.381 to 1.153]
Statistical Analysis 45: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2007637 Genotype: G/A; Test type: Superiority or Other; p = 0.8586, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.114, 95% CI 2-sided [0.339 to 3.667]
Statistical Analysis 46: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2302273 Genotype: G/G; Test type: Superiority or Other; p = 0.8478, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.935, 95% CI 2-sided [0.470 to 1.861]
Statistical Analysis 47: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2302273 Genotype: G/A; Test type: Superiority or Other; p = 0.2445, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.634, 95% CI 2-sided [0.287 to 1.401]
Statistical Analysis 48: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2302273 Genotype: A/A; Test type: Superiority or Other; p = 0.9191, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.155, 95% CI 2-sided [0.072 to 18.59]

50. Secondary Outcome: OS in Subgroups That Were Defined by Germline PDGFRB Polymorphisms
Description: OS, defined as time from date of randomization to date of death due to any cause, in subgroups that were defined by PDGFRB polymorphisms. OS was calculated as (date of death minus date of randomization plus 1) divided by 30.4.
Time Frame: From randomization to Weeks 8 and 12, then every 8 weeks until disease progression or death (up to Month 17)
Population: Per Protocol Caucasian Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 53 | 50
Months
  Locus: PDGFRB/rs2304060 Genotype: C/C | 12.80 [5.60 to 14.00] | 9.60 [4.30 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times
  Locus: PDGFRB/rs2304060 Genotype: C/A | 8.20 [5.40 to 11.30] | 6.20 [4.80 to 14.40]
  Locus: PDGFRB/rs2304060 Genotype: A/A | 5.70 [4.70 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times | 5.60 [3.20 to 16.70]
  Locus: PDGFRB/rs17656204 Genotype: C/C | 8.00 [4.90 to 16.30] | 5.90 [4.40 to 16.70]
  Locus: PDGFRB/rs17656204 Genotype: C/T | 8.20 [5.40 to 11.30] | 7.60 [3.20 to 14.40]
  Locus: PDGFRB/rs17656204 Genotype: T/T | 6.40 [5.60 to 12.80] | NA [4.30 to NA] — Data were not calculable due to the large number of censored event times
  Locus: PDGFRB/rs2304061 Genotype: G/G | 6.65 [5.40 to 11.60] | 4.75 [3.90 to 17.00]
  Locus: PDGFRB/rs2304061 Genotype: G/A | 8.40 [4.20 to 11.30] | 9.60 [5.30 to 14.40]
  Locus: PDGFRB/rs2304061 Genotype: A/A | 9.00 [5.20 to 12.80] | NA [NA to NA] — Number of participants in this category was zero
  Locus: PDGFRB/rs1077724 Genotype: A/A | 6.30 [4.90 to 11.60] | 5.90 [4.40 to 16.70]
  Locus: PDGFRB/rs1077724 Genotype: A/T | 9.70 [6.40 to 14.00] | 6.20 [4.20 to 14.40]
  Locus: PDGFRB/rs1077724 Genotype: T/T | 7.25 [3.10 to 12.80] | NA [7.20 to NA] — Data were not calculable due to the large number of censored event times
  Locus: PDGFRB/rs919751 Genotype: A/A | 8.00 [5.10 to 14.00] | 6.80 [4.20 to 13.40]
  Locus: PDGFRB/rs919751 Genotype: A/G | 8.20 [6.20 to 11.30] | 10.00 [4.40 to 16.50]
  Locus: PDGFRB/rs919751 Genotype: G/G | 6.40 [1.80 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times | 8.20 [2.20 to 17.20]
  Locus: PDGFRB/rs2304058 Genotype: G/G | 6.05 [4.70 to 9.30] | 8.45 [4.40 to 17.00]
  Locus: PDGFRB/rs2304058 Genotype: G/C | 8.20 [5.60 to 11.60] | 7.20 [4.20 to 14.40]
  Locus: PDGFRB/rs2304058 Genotype: C/C | 12.05 [8.00 to 14.00] | 6.20 [4.60 to 13.40]
  Locus: PDGFRB/rs1864972 Genotype: G/G | 6.65 [5.10 to 11.60] | 11.50 [4.40 to 17.00]
  Locus: PDGFRB/rs1864972 Genotype: G/A | 8.00 [5.60 to 11.30] | 6.35 [4.20 to 14.40]
  Locus: PDGFRB/rs1864972 Genotype: A/A | 11.30 [4.10 to 12.80] | 7.90 [3.20 to 13.40]
  Locus: PDGFRB/rs3733678 Genotype: G/G | 6.30 [5.20 to 9.30] | 7.00 [4.40 to 13.40]
  Locus: PDGFRB/rs3733678 Genotype: G/A | 14.00 [11.6 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times | 5.90 [4.40 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times
  Locus: PDGFRB/rs246396 Genotype: T/T | 8.00 [5.70 to 16.30] | 5.40 [4.30 to 10.00]
  Locus: PDGFRB/rs246396 Genotype: T/C | 7.30 [4.10 to 11.30] | 14.95 [7.20 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times
  Locus: PDGFRB/rs246396 Genotype: C/C | NA [NA to NA] — Number of participants in this category was zero | 6.20 [NA to NA] — Number of participants in this category was 1
  Locus: PDGFRB/rs34586048 Genotype: C/C | 8.00 [5.70 to 11.30] | 6.80 [4.80 to 13.40]
  Locus: PDGFRB/rs11740355 Genotype: T/T | 8.20 [5.60 to 11.30] | 6.20 [4.60 to 11.50]
  Locus: PDGFRB/rs11740355 Genotype: T/G | 6.90 [4.70 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times | 14.40 [2.20 to 17.00]
  Locus: PDGFRB/rs11740355 Genotype: G/G | 1.80 [NA to NA] — Number of participants in this category was 1 | NA [NA to NA] — Number of participants in this category was zero
  Locus: PDGFRB/rs740751 Genotype: C/C | 6.65 [5.10 to 11.60] | 11.50 [4.40 to 17.00]
  Locus: PDGFRB/rs740751 Genotype: C/T | 8.00 [5.60 to 11.30] | 6.80 [4.30 to 14.40]
  Locus: PDGFRB/rs740751 Genotype: T/T | 11.30 [4.10 to 12.80] | 7.90 [3.20 to 13.40]
  Locus: PDGFRB/rs4705415 Genotype: G/G | 11.30 [8.00 to 14.00] | 6.70 [4.60 to 13.40]
  Locus: PDGFRB/rs4705415 Genotype: G/A | 8.20 [5.60 to 11.30] | 6.80 [4.30 to 17.00]
  Locus: PDGFRB/rs4705415 Genotype: A/A | 5.60 [3.70 to 6.90] | 8.20 [2.20 to 17.20]
  Locus: PDGFRB/rs3776075 Genotype: T/T | 6.35 [4.70 to 8.40] | 14.35 [2.20 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times
  Locus: PDGFRB/rs3776075 Genotype: T/G | 9.30 [5.20 to 11.30] | 7.20 [4.90 to 16.50]
  Locus: PDGFRB/rs3776075 Genotype: G/G | 14.00 [4.80 to 16.30] | 4.70 [3.20 to 7.60]
  Locus: PDGFRB/rs17708574 Genotype: G/G | 9.30 [6.40 to 11.60] | 6.20 [4.60 to 13.40]
  Locus: PDGFRB/rs17708574 Genotype: G/A | 5.40 [4.20 to 6.30] | 6.80 [3.90 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times
  Locus: PDGFRB/rs10063714 Genotype: T/T | 6.40 [5.40 to 9.30] | 7.20 [4.80 to 14.40]
  Locus: PDGFRB/rs10063714 Genotype: T/A | 14.00 [11.6 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times | 5.90 [3.90 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times
  Locus: PDGFRB/rs3776081 Genotype: A/A | 6.30 [5.10 to 8.40] | 12.95 [4.90 to 17.20]
  Locus: PDGFRB/rs3776081 Genotype: A/G | 11.30 [5.70 to 12.80] | 6.80 [4.20 to 13.40]
  Locus: PDGFRB/rs3776081 Genotype: G/G | 11.60 [4.80 to 14.00] | 4.80 [3.20 to 9.60]
  Locus: PDGFRB/rs2007637 Genotype: G/G | 6.90 [5.40 to 11.60] | 5.40 [4.30 to 10.00]
  Locus: PDGFRB/rs2007637 Genotype: G/A | 8.20 [5.60 to 9.30] | 13.40 [7.20 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times
  Locus: PDGFRB/rs2007637 Genotype: A/A | 8.40 [NA to NA] — Number of participants in this category was 1 | NA [NA to NA] — Number of participants in this category was zero
  Locus: PDGFRB/rs2302273 Genotype: G/G | 7.55 [5.60 to 9.70] | 11.50 [4.90 to 17.20]
  Locus: PDGFRB/rs2302273 Genotype: G/A | 11.30 [5.70 to 12.80] | 6.20 [3.90 to 13.40]
  Locus: PDGFRB/rs2302273 Genotype: A/A | 4.80 [4.10 to NA] — Upper limit of confidence interval was not calculable due to the large number of censored event times | 4.80 [1.10 to 9.60]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2304060 Genotype: C/C; Test type: Superiority or Other; p = 0.8563, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.121, 95% CI 2-sided [0.326 to 3.847]
Statistical Analysis 2: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2304060 Genotype: C/A; Test type: Superiority or Other; p = 0.7375, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.111, 95% CI 2-sided [0.599 to 2.064]
Statistical Analysis 3: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs234060 Genotype: A/A; Test type: Superiority or Other; p = 0.8066, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.897, 95% CI 2-sided [0.375 to 2.147]
Statistical Analysis 4: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs17656204 Genotype: C/C; Test type: Superiority or Other; p = 0.6945, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.875, 95% CI 2-sided [0.449 to 1.708]
Statistical Analysis 5: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs17656204 Genotype: C/T; Test type: Superiority or Other; p = 0.8536, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.067, 95% CI 2-sided [0.536 to 2.122]
Statistical Analysis 6: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs17656204 Genotype: T/T; Test type: Superiority or Other; p = 0.3657, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 2.732, 95% CI 2-sided [0.283 to 26.42]
Statistical Analysis 7: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2304061 Genotype: G/G; Test type: Superiority or Other; p = 0.4657, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.793, 95% CI 2-sided [0.424 to 1.483]
Statistical Analysis 8: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2304061 Genotype: G/A; Test type: Superiority or Other; p = 0.4168, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.364, 95% CI 2-sided [0.641 to 2.900]
Statistical Analysis 9: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs1077724 Genotype: A/A; Test type: Superiority or Other; p = 0.7836, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.908, 95% CI 2-sided [0.456 to 1.809]
Statistical Analysis 10: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs1077724 Genotype: A/T; Test type: Superiority or Other; p = 0.8531, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.938, 95% CI 2-sided [0.472 to 1.863]
Statistical Analysis 11: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs1077724 Genotype: T/T; Test type: Superiority or Other; p = 0.3272, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 2.320, 95% CI 2-sided [0.412 to 13.07]
Statistical Analysis 12: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs919751 Genotype: A/A; Test type: Superiority or Other; p = 0.9630, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.984, 95% CI 2-sided [0.491 to 1.972]
Statistical Analysis 13: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs919751 Genotype: A/G; Test type: Superiority or Other; p = 0.6003, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.227, 95% CI 2-sided [0.567 to 2.656]
Statistical Analysis 14: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs919751 Genotype: G/G; Test type: Superiority or Other; p = 0.6703, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.769, 95% CI 2-sided [0.229 to 2.580]
Statistical Analysis 15: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2304058 Genotype: G/G; Test type: Superiority or Other; p = 0.8100, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.106, 95% CI 2-sided [0.485 to 2.525]
Statistical Analysis 16: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2304058 Genotype: G/C; Test type: Superiority or Other; p = 0.8335, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.076, 95% CI 2-sided [0.541 to 2.141]
Statistical Analysis 17: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2304058 Genotype: C/C; Test type: Superiority or Other; p = 0.5980, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.758, 95% CI 2-sided [0.268 to 2.141]
Statistical Analysis 18: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs1864972 Genotype: G/G; Test type: Superiority or Other; p = 0.9287, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.035, 95% CI 2-sided [0.487 to 2.199]
Statistical Analysis 19: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs1864972 Genotype: G/A; Test type: Superiority or Other; p = 0.8842, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.053, 95% CI 2-sided [0.526 to 2.106]
Statistical Analysis 20: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs1864972 Genotype: A/A; Test type: Superiority or Other; p = 0.8501, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.129, 95% CI 2-sided [0.316 to 4.028]
Statistical Analysis 21: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs3733678 Genotype: G/G; Test type: Superiority or Other; p = 0.4118, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.229, 95% CI 2-sided [0.749 to 2.017]
Statistical Analysis 22: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs3733678 Genotype: G/A; Test type: Superiority or Other; p = 0.1299, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.286, 95% CI 2-sided [0.051 to 1.596]
Statistical Analysis 23: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs246396 Genotype: T/T; Test type: Superiority or Other; p = 0.1859, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.692, 95% CI 2-sided [0.399 to 1.200]
Statistical Analysis 24: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs246396 Genotype: T/C; Test type: Superiority or Other; p = 0.0091, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 3.672, 95% CI 2-sided [1.291 to 10.44]
Statistical Analysis 25: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs34586048 Genotype: C/C; Test type: Superiority or Other; p = 0.8708, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.039, 95% CI 2-sided [0.654 to 1.652]
Statistical Analysis 26: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs11740355 Genotype: T/T; Test type: Superiority or Other; p = 0.9888, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.996, 95% CI 2-sided [0.590 to 1.681]
Statistical Analysis 27: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs11740355 Genotype: T/G; Test type: Superiority or Other; p = 0.9702, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.020, 95% CI 2-sided [0.360 to 2.891]
Statistical Analysis 28: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs740751 Genotype: C/C; Test type: Superiority or Other; p = 0.9419, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.973, 95% CI 2-sided [0.466 to 2.032]
Statistical Analysis 29: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs740751 Genotype: C/T; Test type: Superiority or Other; p = 0.7677, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.112, 95% CI 2-sided [0.549 to 2.252]
Statistical Analysis 30: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs740751 Genotype: T/T; Test type: Superiority or Other; p = 0.8501, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.129, 95% CI 2-sided [0.316 to 4.028]
Statistical Analysis 31: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs4705415 Genotype: G/G; Test type: Superiority or Other; p = 0.5233, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.758, 95% CI 2-sided [0.322 to 1.782]
Statistical Analysis 32: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs4705415 Genotype: G/A; Test type: Superiority or Other; p = 0.7500, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.123, 95% CI 2-sided [0.549 to 2.297]
Statistical Analysis 33: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs4705415 Genotype: A/A; Test type: Superiority or Other; p = 0.6614, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.232, 95% CI 2-sided [0.483 to 3.142]
Statistical Analysis 34: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs3776075 Genotype: T/T; Test type: Superiority or Other; p = 0.2552, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.779, 95% CI 2-sided [0.652 to 4.855]
Statistical Analysis 35: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs3776075 Genotype: T/G; Test type: Superiority or Other; p = 0.7931, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.088, 95% CI 2-sided [0.577 to 2.052]
Statistical Analysis 36: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs3776075 Genotype: G/G; Test type: Superiority or Other; p = 0.1365, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.449, 95% CI 2-sided [0.152 to 1.331]
Statistical Analysis 37: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs17708574 Genotype: G/G; Test type: Superiority or Other; p = 0.5544, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.854, 95% CI 2-sided [0.504 to 1.447]
Statistical Analysis 38: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs17708574 Genotype: G/A; Test type: Superiority or Other; p = 0.3132, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.721, 95% CI 2-sided [0.590 to 5.021]
Statistical Analysis 39: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs10063714 Genotype: T/T; Test type: Superiority or Other; p = 0.3698, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.263, 95% CI 2-sided [0.755 to 2.113]
Statistical Analysis 40: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs10063714 Genotype: T/A; Test type: Superiority or Other; p = 0.1495, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.411, 95% CI 2-sided [0.119 to 1.423]
Statistical Analysis 41: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs3776081 Genotype: A/A; Test type: Superiority or Other; p = 0.1911, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.613, 95% CI 2-sided [0.781 to 3.332]
Statistical Analysis 42: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs3776081 Genotype: A/G; Test type: Superiority or Other; p = 0.5259, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.793, 95% CI 2-sided [0.384 to 1.636]
Statistical Analysis 43: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs3776081 Genotype: G/G; Test type: Superiority or Other; p = 0.0996, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.331, 95% CI 2-sided [0.082 to 1.339]
Statistical Analysis 44: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2007637 Genotype: G/G; Test type: Superiority or Other; p = 0.2755, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.752, 95% CI 2-sided [0.450 to 1.259]
Statistical Analysis 45: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2007637 Genotype: G/A; Test type: Superiority or Other; p = 0.0120, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 4.850, 95% CI 2-sided [1.253 to 18.78]
Statistical Analysis 46: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2302273 Genotype: G/G; Test type: Superiority or Other; p = 0.4663, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 1.274, 95% CI 2-sided [0.661 to 2.457]
Statistical Analysis 47: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2302273 Genotype: G/A; Test type: Superiority or Other; p = 0.7097, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.867, 95% CI 2-sided [0.406 to 1.848]
Statistical Analysis 48: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Locus: PDGFRB/rs2302273 Genotype: A/A; Test type: Superiority or Other; p = 0.5340, Log Rank — 2-sided unstratified log-rank test; Hazard Ratio (HR) = 0.607, 95% CI 2-sided [0.117 to 3.158]

51. Secondary Outcome: Percentage of Participants by Tumor VEGFR Mutation
Description: Percentage of participants with VEGFR mutations in DNA from tumor samples collected at the time of initial diagnosis (preferred) or at the time of most recent recurrence/progression, although any time was acceptable.
Time Frame: Baseline
Population: Full Analysis - All Population; data were not analyzed
Arm/Group | All Participants
Number analyzed (Participants) | 0

52. Secondary Outcome: Correlation of Polymorphisms in Stem Cell Factor Receptor (c-Kit), FMS-like Tyrosine Kinase 3 Receptor (FLT-3), and c-FMS With Blood Counts
Description: A blood sample (6 mL) was collected before on-study treatment and was used to isolate DNA. These samples were not anonymized. Correlation was investigated by the percentage of participants with anemia (based on hemoglobin count), neutropenia (based on neutrophil count) and thrombocytopenia (based on platelet count) endpoints and genetic variation as measured by c-KIT, FLT-3, and c-FMS was to be analyzed.
Time Frame: Baseline (Day 1, Cycle 1)
Population: Blood samples were collected; however, because of the small sample size that resulted in a lack of power for statistical testing, no formal statistical analyses were performed.
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 0 | 0

53. Other Pre Specified Outcome: VEGF-C Ratio to Baseline at Each Timepoint
Description: Plasma VEGF-C concentration at each time point divided by VEGF-C concentration at baseline (ratio to baseline)
Time Frame: Baseline to Cycle 2 (Day 1) and Cycle 3 (Day 1)
Population: FA Set; n equals number of participants with evaluable data at specified cycle
Measure: Median (Full Range); unit: Ratio
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Ratio
  Cycle 2, Day 1 (n=41, 46) | 0.86 [0.29 to 2.40] | 1.02 [0.32 to 2.86]
  Cycle 3, Day 1 (n=36, 35) | 0.95 [0.15 to 2.53] | 0.95 [0.20 to 4.91]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; VEGF-C Ratio to Baseline for Cycle 2, Day 1; Test type: Superiority or Other; p = 0.2702, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; VEGF-C ratio to Baseline for Cycle 3, Day 1; Test type: Superiority or Other; p = 0.7354, Wilcoxon Rank Sum Test

54. Secondary Outcome: Percentage of Participants by Ribonucleic Acid (RNA) Expression Profile
Description: Includes colony-stimulating factor 1 receptor (CSF-1R), PDGFRalpha, PDGFRbeta, vascular endothelial growth factor (VEGF), VEGF C (VEGF-C), VEGF receptor 1 (VEGFR1), VEGF receptor 2 (VEGFR2), VEGF receptor 3 (VEGFR3), fibroblast growth factor (FGF), FLT-3, KIT (stem cell factor receptor), and RET (rearranged during transfection). Correlative analysis was conducted using tumor biopsy samples collected at the time of initial diagnosis (preferred) or at the time of most recent recurrence/progression, although any time was acceptable.
Time Frame: Baseline
Population: FA Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Percentage of Participants
  CSF-1R/High | 45 | 44
  CSF-1R/Low | 52 | 41
  CSF-1R/Indeterminate | 3 | 15
  PDGFRalpha/High | 45 | 48
  PDGFRalpha/Low | 52 | 41
  PDGFRalpha/Indeterminate | 3 | 11
  PDGFRbeta/High | 45 | 44
  PDGFRbeta/Low | 48 | 44
  PDGFRbeta/Indeterminate | 6 | 11
  VEGF/High | 39 | 41
  VEGF/Low | 39 | 41
  VEGF/Indeterminate | 23 | 19
  VEGF-C/High | 52 | 41
  VEGF-C/Low | 45 | 52
  VEGF-C/Indeterminate | 3 | 7
  VEGFR1/High | 35 | 44
  VEGFR1/Low | 48 | 33
  VEGFR1/Indeterminate | 16 | 22
  VEGFR2/High | 45 | 48
  VEGFR2/Low | 52 | 41
  VEGFR2/Indeterminate | 3 | 11
  VEGFR3/High | 35 | 48
  VEGFR3/Low | 55 | 30
  VEGFR3/Indeterminate | 10 | 22
  FGF/Detected | 10 | 19
  FGF/Not Detected | 84 | 67
  FGF/Indeterminate | 6 | 15
  FLT3/Detected | 26 | 19
  FLT3/Not Detected | 71 | 78
  FLT3/Indeterminate | 3 | 4
  KIT/Detected | 39 | 30
  KIT/Not Detected | 58 | 67
  KIT/Indeterminate | 3 | 4
  RET/Detected | 10 | 30
  RET/Not Detected | 84 | 59
  RET/Indeterminate | 6 | 11

55. Other Pre Specified Outcome: VEGFR-2 Ratio to Baseline at Each Timepoint
Description: Plasma VEGFR-2 concentration at each time point divided by VEGFR-2 concentration at baseline (ratio to baseline)
Time Frame: Baseline to Cycle 2 (Day 1) and Cycle 3 (Day 1)
Population: FA Set; n equals number of participants with evaluable data at specified cycle
Measure: Median (Full Range); unit: Ratio
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Ratio
  Cycle 2, Day 1 (n=43, 46) | 0.71 [0.40 to 1.36] | 0.98 [0.63 to 1.66]
  Cycle 3, Day 1 (n=36, 36) | 0.67 [0.43 to 1.02] | 0.99 [0.64 to 1.78]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; VEGFR-2 Ratio to Baseline for Cycle 2, Day 1; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; VEGFR-2 Ratio to Baseline for Cycle 3, Day 1; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum Test

56. Secondary Outcome: PFS in Subgroups That Were Defined by RNA Expression Profile
Description: PFS, defined as time from date of randomization to date of first documentation of PD or death on-study due to any cause, whichever occurred first, in subgroups that were defined by RNA Gene expression (CSF-1R, PDGFRalpha, PDGFRbeta, VEGF, VEGF-C, VEGFR1, VEGFR2, VEGFR3, FGF, FLT-3, KIT, and RET). PFS was calculated as (first event date minus randomization date plus 1) divided by 7.02.
Time Frame: From randomization to Weeks 8 and 12, then every 8 weeks until disease progression or death (up to Month 17)
Population: FA Set
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Weeks
  CSF-1R/High | 19.1 [9.00 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times | 10.9 [7.70 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times
  CSF-1R/Low | 12.3 [7.80 to 19.50] | 12.3 [7.50 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times
  CSF-1R/Indeterminate | 9.5 [5.30 to 20.70] | 8.1 [7.70 to 12.80]
  PDGFRalpha/High | 12.3 [8.10 to 19.10] | 52.0 [10.10 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times
  PDGFRalpha/Low | 16.0 [7.80 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times | 7.7 [7.10 to 11.70]
  PDGFRalpha/Indeterminate | 9.5 [5.30 to 20.70] | 8.1 [7.80 to 12.80]
  PDGFRbeta/High | 12.3 [8.10 to 20.10] | 11.7 [7.50 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times
  PDGFRbeta/Low | 16.0 [7.80 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times | 12.3 [8.80 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times
  PDGFRbeta/Indeterminate | 9.5 [5.40 to 20.50] | 8.1 [7.80 to 12.80]
  VEGF/High | 16.0 [8.10 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times | 10.1 [7.70 to 52.00]
  VEGF/Low | 19.1 [7.80 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times | 11.7 [7.50 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times
  VEGF/Indeterminate | 9.5 [7.70 to 20.10] | 8.1 [7.80 to 12.80]
  VEGF-C/High | 12.3 [8.10 to 20.10] | 12.1 [10.10 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times
  VEGF-C/Low | 16.0 [7.80 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times | 8.5 [7.50 to 52.0]
  VEGF-C/Indeterminate | 9.5 [5.30 to 20.70] | 8.1 [7.70 to 12.80]
  VEGFR1/High | 12.5 [8.10 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times | 11.2 [7.70 to 52.00]
  VEGFR1/Low | 19.1 [7.80 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times | 11.7 [8.80 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times
  VEGFR1/Indeterminate | 9.5 [7.70 to 20.10] | 8.1 [7.70 to 12.30]
  VEGFR2/High | 17.0 [9.00 to 20.10] | 12.3 [7.70 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times
  VEGFR2/Low | 16.0 [7.80 to 19.10] | 8.8 [5.40 to 52.00]
  VEGFR2/Indeterminate | 9.5 [5.30 to 20.70] | 8.1 [7.80 to 12.80]
  VEGFR3/High | NA [8.10 to NA] — data were not calculable due to the large number of censored event times | 12.3 [8.50 to 52.00]
  VEGFR3/Low | 12.3 [7.80 to 19.10] | 8.8 [5.40 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times
  VEGFR3/Indeterminate | 9.5 [5.40 to 20.50] | 8.0 [7.70 to 12.30]
  FGF/Detected | 11.7 [7.40 to 16.00] | 7.7 [4.80 to 10.10]
  FGF/Not Detected | 12.3 [8.10 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times | 12.3 [8.80 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times
  FGF/Indeterminate | 9.5 [5.40 to 20.50] | 8.1 [7.70 to 12.30]
  FLT3/Detected | 16.0 [9.00 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times | 12.1 [11.70 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times
  FLT3/Not Detected | 17.0 [7.80 to 20.10] | 8.5 [7.50 to 52.00]
  FLT3/Indeterminate | 9.5 [5.30 to 20.70] | 8.1 [7.80 to 12.80]
  KIT/Detected | 19.5 [7.40 to 20.10] | 10.1 [8.50 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times
  KIT/Not Detected | 16.0 [9.00 to 19.10] | 11.7 [7.50 to 52.00]
  KIT/Indeterminate | 9.5 [5.30 to 20.70] | 8.1 [7.80 to 12.80]
  RET/Detected | 10.4 [4.70 to 16.00] | 10.1 [8.50 to 12.30]
  RET/Not Detected | 12.3 [8.10 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times | 11.7 [7.50 to NA] — upper limit of confidence interval was not calculable due to the large number of censored event times
  RET/Indeterminate | 9.5 [5.40 to 20.50] | 8.1 [7.80 to 12.80]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; High CSF-1R expression; Test type: Superiority or Other; p = 0.1667, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.553, 95% CI 2-sided [0.159 to 1.921]
Statistical Analysis 2: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Low CSF-1R expression; Test type: Superiority or Other; p = 0.7688, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 1.451, 95% CI 2-sided [0.534 to 3.944]
Statistical Analysis 3: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Indeterminate CSF-1R expression; Test type: Superiority or Other; p = 0.3498, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.890, 95% CI 2-sided [0.503 to 1.574]
Statistical Analysis 4: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; High PDGFRalpha expression; Test type: Superiority or Other; p = 0.9497, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 2.687, 95% CI 2-sided [0.790 to 9.143]
Statistical Analysis 5: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Low PDGFRalpha expression; Test type: Superiority or Other; p = 0.0401, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.386, 95% CI 2-sided [0.127 to 1.173]
Statistical Analysis 6: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Indeterminate PDGFRalpha expression; Test type: Superiority or Other; p = 0.3128, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.862, 95% CI 2-sided [0.487 to 1.524]
Statistical Analysis 7: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; High PDGFRbeta expression; Test type: Superiority or Other; p = 0.3650, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.823, 95% CI 2-sided [0.273 to 2.488]
Statistical Analysis 8: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Low PDGFRbeta expression; Test type: Superiority or Other; p = 0.6105, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 1.192, 95% CI 2-sided [0.408 to 3.480]
Statistical Analysis 9: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Indeterminate PDGFRbeta expression; Test type: Superiority or Other; p = 0.3027, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.856, 95% CI 2-sided [0.488 to 1.502]
Statistical Analysis 10: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; High VEGF expression; Test type: Superiority or Other; p = 0.4436, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.914, 95% CI 2-sided [0.262 to 3.184]
Statistical Analysis 11: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Low VEGF expression; Test type: Superiority or Other; p = 0.4582, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.953, 95% CI 2-sided [0.296 to 3.062]
Statistical Analysis 12: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Indeterminate VEGF expression; Test type: Superiority or Other; p = 0.3720, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.911, 95% CI 2-sided [0.536 to 1.548]
Statistical Analysis 13: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; High VEGF-C expression; Test type: Superiority or Other; p = 0.5586, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 1.090, 95% CI 2-sided [0.350 to 3.397]
Statistical Analysis 14: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Low VEGF-C expression; Test type: Superiority or Other; p = 0.3652, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.842, 95% CI 2-sided [0.313 to 2.266]
Statistical Analysis 15: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Indeterminate VEGF-C expression; Test type: Superiority or Other; p = 0.3301, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.875, 95% CI 2-sided [0.493 to 1.554]
Statistical Analysis 16: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; High VEGFR1 expression; Test type: Superiority or Other; p = 0.5605, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 1.097, 95% CI 2-sided [0.331 to 3.636]
Statistical Analysis 17: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Low VEGFR1 expression; Test type: Superiority or Other; p = 0.2132, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.599, 95% CI 2-sided [0.160 to 2.236]
Statistical Analysis 18: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Indeterminate VEGFR1 expression; Test type: Superiority or Other; p = 0.3605, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.902, 95% CI 2-sided [0.530 to 1.537]
Statistical Analysis 19: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; High VEGFR2 expression; Test type: Superiority or Other; p = 0.4438, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.921, 95% CI 2-sided [0.304 to 2.784]
Statistical Analysis 20: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Low VEGFR2 expression; Test type: Superiority or Other; p = 0.5699, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 1.122, 95% CI 2-sided [0.403 to 3.125]
Statistical Analysis 21: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Indeterminate VEGFR2 expression; Test type: Superiority or Other; p = 0.3147, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.864, 95% CI 2-sided [0.489 to 1.528]
Statistical Analysis 22: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; High VEGFR3 expression; Test type: Superiority or Other; p = 0.5015, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 1.002, 95% CI 2-sided [0.281 to 3.581]
Statistical Analysis 23: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Low VEGFR3 expression; Test type: Superiority or Other; p = 0.4887, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 1.005, 95% CI 2-sided [0.334 to 3.025]
Statistical Analysis 24: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Indeterminate VEGFR3 expression; Test type: Superiority or Other; p = 0.2432, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.818, 95% CI 2-sided [0.473 to 1.414]
Statistical Analysis 25: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Detected FGF expression; Test type: Superiority or Other; p = 0.2321, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.446, 95% CI 2-sided [0.048 to 4.101]
Statistical Analysis 26: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; No detected FGF expression; Test type: Superiority or Other; p = 0.7143, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 1.316, 95% CI 2-sided [0.526 to 3.292]
Statistical Analysis 27: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Indeterminate FGF expression; Test type: Superiority or Other; p = 0.2812, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.844, 95% CI 2-sided [0.486 to 1.465]
Statistical Analysis 28: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Detected FLT3 expression; Test type: Superiority or Other; p = 0.6504, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 1.406, 95% CI 2-sided [0.248 to 7.960]
Statistical Analysis 29: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; No detected FLT3 expression; Test type: Superiority or Other; p = 0.3266, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.838, 95% CI 2-sided [0.375 to 1.876]
Statistical Analysis 30: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Indeterminate FLT3 expression; Test type: Superiority or Other; p = 0.3597, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.896, 95% CI 2-sided [0.502 to 1.598]
Statistical Analysis 31: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Detected KIT expression; Test type: Superiority or Other; p = 0.6907, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 1.342, 95% CI 2-sided [0.419 to 4.297]
Statistical Analysis 32: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Participants with no detected KIT expression; Test type: Superiority or Other; p = 0.1990, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.677, 95% CI 2-sided [0.265 to 1.731]
Statistical Analysis 33: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Indeterminate KIT expression; Test type: Superiority or Other; p = 0.3597, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.896, 95% CI 2-sided [0.502 to 1.598]
Statistical Analysis 34: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Detected RET expression; Test type: Superiority or Other; p = 0.3757, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.693, 95% CI 2-sided [0.071 to 6.765]
Statistical Analysis 35: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; No detected RET expression; Test type: Superiority or Other; p = 0.3723, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.874, 95% CI 2-sided [0.358 to 2.130]
Statistical Analysis 36: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Indeterminate RET expression; Test type: Superiority or Other; p = 0.3263, Log Rank — 1-sided unstratified log-rank test; Hazard Ratio (HR) = 0.874, 95% CI 2-sided [0.501 to 1.523]

57. Other Pre Specified Outcome: VEGFR-3 Ratio to Baseline at Each Timepoint
Description: Plasma VEGFR-3 concentration at each time point divided by VEGFR-3 concentration at baseline (ratio to baseline)
Time Frame: Baseline to Cycle 2 (Day 1) and Cycle 3 (Day 1)
Population: FA Set; n equals number of participants with evaluable data at specified cycle
Measure: Median (Full Range); unit: Ratio
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Ratio
  Cycle 2, Day 1 (n=43, 47) | 0.60 [0.29 to 1.28] | 0.98 [0.48 to 2.37]
  Cycle 3, Day 1 (n=36, 36) | 0.57 [0.31 to 1.37] | 0.92 [0.60 to 2.04]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; VEGFR-3 Ratio to Baseline for Cycle 2, Day 1; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; VEGFR-3 Ratio to Baseline for Cycle 3, Day 1; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum Test

58. Secondary Outcome: Health Related Quality of Life (HRQoL) and Lung Cancer Related Symptoms as Assessed With European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) Score
Description: EORTC QLQ-C30: self-administered questionnaire assessing global health status/quality of life (QoL), functional domains (physical, role, cognitive, emotional, and social), symptom scales/items (fatigue, pain, nausea and vomiting, dyspnea, insomnia, loss of appetite, constipation, and diarrhea), and financial difficulties. Recall period: past week; response range: not at all (1) to very much (4); global/QoL range: very poor (1) to excellent (7). Scale score range: 0 to 100. Higher functional/global QoL score = better functioning and higher symptom score = greater degree of symptoms.
Time Frame: Baseline (Cycle [C] 1, Day [D] 1) to Cycle 18, Day 1
Population: Patient-Reported Outcome (PRO) Analysis Set: participants from the FA Set who had at least 1 EORTC QLQ-C30 or EORTC QLQ Lung cancer (QLQ-LC13) module questionnaire assessment while on treatment; n is number of participants with an assessment at the specified time point.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 49 | 54
score on a scale
  Global Health Status/QoL (C1, D1) (n=49, 53) | 66.49 [59.75 to 73.24] | 62.26 [56.81 to 67.71]
  Global Health Status/QoL (C2, D1) (n=41, 46) | 62.60 [55.47 to 69.74] | 57.43 [50.28 to 64.59]
  Global Health Status/QoL (C3, D1) (n=27, 32) | 61.73 [52.18 to 71.29] | 59.12 [50.47 to 67.77]
  Global Health Status/QoL (C4, D1) (n=19, 22) | 66.67 [55.47 to 77.86] | 60.98 [51.28 to 70.68]
  Global Health Status/QoL (C5, D1) (n=14, 18) | 69.05 [55.92 to 82.18] | 61.12 [50.88 to 71.37]
  Global Health Status/QoL (C6, D1) (n=8, 14) | 80.20 [65.80 to 94.60] | 67.27 [59.62 to 74.93]
  Global Health Status/QoL (C7, D1) (n=7, 10) | 71.41 [54.85 to 87.98] | 63.34 [48.42 to 78.26]
  Global Health Status/QoL (C8, D1) (n=4, 7) | 89.60 [64.52 to 100.00] | 59.51 [34.97 to 84.06]
  Global Health Status/QoL (C9, D1) (n=4, 5) | 79.18 [39.40 to 100.00] | 66.66 [37.40 to 95.92]
  Global Health Status/QoL (C10, D1) (n=3, 4) | 88.90 [41.14 to 100.00] | 56.25 [16.61 to 95.89]
  Global Health Status/QoL (C11, D1) (n=3, 4) | 86.10 [54.47 to 100.00] | 62.50 [22.72 to 100.00]
  Global Health Status/QoL (C12, D1) (n=3, 4) | 88.90 [57.27 to 100.00] | 58.33 [31.83 to 84.82]
  Global Health Status/QoL (C13, D1) (n=3, 3) | 80.57 [0.00 to 100.00] | 61.10 [13.34 to 100.00]
  Global Health Status/QoL (C14, D1) (n=2, 3) | 75.00 [0.00 to 100.00] | 55.53 [0.00 to 100.00]
  Global Health Status/QoL (C15, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | 66.65 [0.00 to 100.00]
  Global Health Status/QoL (C16, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | 66.65 [0 to 100.00]
  Global Health Status/QoL (C17, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | 58.30 [0 to 100.00]
  Global Health Status/QoL (C18, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | 66.65 [0 to 100.00]
  Physical Functioning (C1, D1) (n=49, 54) | 79.32 [74.36 to 84.29] | 74.81 [69.13 to 80.50]
  Physical Functioning (C2, D1) (n=41, 46) | 77.24 [70.99 to 83.48] | 72.03 [65.21 to 78.86]
  Physical Functioning (C3, D1) (n=28, 32) | 73.58 [65.79 to 81.37] | 72.28 [65.11 to 79.46]
  Physical Functioning (C4, D1) (n=19, 22) | 71.58 [60.41 to 82.76] | 74.23 [64.48 to 83.99]
  Physical Functioning (C5, D1) (n=14, 18) | 75.72 [60.21 to 91.24] | 68.89 [57.81 to 79.97]
  Physical Functioning (C6, D1) (n=9, 14) | 85.92 [74.05 to 97.80] | 75.24 [63.60 to 86.87]
  Physical Functioning (C7, D1) (n=7, 10) | 80.00 [58.05 to 100.00] | 71.99 [58.54 to 85.44]
  Physical Functioning (C8, D1) (n=4, 7) | 93.35 [81.13 to 100.00] | 74.29 [54.66 to 93.91]
  Physical Functioning (C9, D1) (n=4, 5) | 95.00 [84.86 to 100.00] | 73.32 [44.07 to 100.00]
  Physical Functioning (C10, D1) (n=3, 4) | 93.33 [64.65 to 100.00] | 70.00 [39.43 to 100.00]
  Physical Functioning (C11, D1) (n=3, 4) | 93.33 [76.81 to 100.00] | 71.68 [40.04 to 100.00]
  Physical Functioning (C12, D1) (n=3, 4) | 97.77 [88.16 to 100.00] | 71.68 [40.04 to 100.00]
  Physical Functioning (C13, D1) (n=3, 3) | 95.57 [76.49 to 100.00] | 73.30 [23.62 to 100.00]
  Physical Functioning (C14, D1) (n=2, 3) | 93.35 [8.85 to 100.00] | 68.90 [10.83 to 100.00]
  Physical Functioning (C15, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | 70.00 [0 to 100.00]
  Physical Functioning (C16, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | 66.70 [0 to 100.00]
  Physical Functioning (C17, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | 70.00 [0 to 100.00]
  Physical Functioning (C18, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | 73.30 [0 to 100.00]
  Role Functioning (C1, D1) (n=49, 53) | 80.95 [73.97 to 87.93] | 69.18 [60.52 to 77.84]
  Role Functioning (C2, D1) (n=41, 46) | 67.89 [57.68 to 78.11] | 64.13 [54.52 to 73.75]
  Role Functioning (C3, D1) (n=28, 32) | 72.63 [61.90 to 83.35] | 64.07 [52.13 to 76.00]
  Role Functioning (C4, D1) (n=19, 22) | 68.43 [55.06 to 81.79] | 67.43 [55.04 to 79.81]
  Role Functioning (C5, D1) (n=14, 17) | 69.06 [51.83 to 86.30] | 67.65 [53.94 to 81.35]
  Role Functioning (C6, D1) (n=9, 14) | 83.34 [67.66 to 99.03] | 69.05 [49.86 to 88.24]
  Role Functioning (C7, D1) (n=7,10) | 85.71 [66.99 to 100.00] | 73.34 [60.53 to 86.15]
  Role Functioning (C8, D1) (n=4, 7) | 91.68 [65.18 to 100.00] | 69.04 [38.97 to 99.12]
  Role Functioning (C9, D1) (n=4, 5) | 91.68 [65.18 to 100.00] | 66.66 [25.25 to 100.00]
  Role Functioning (C10, D1) (n=3, 4) | 94.43 [70.48 to 100.00] | 50.00 [0 to 100.00]
  Role Functioning (C11, D1) (n=3, 4) | 94.43 [70.48 to 100.00] | 62.50 [17.19 to 100.00]
  Role Functioning (C12, D1) (n=3, 4) | 100.00 [100.00 to 100.00] | 62.50 [17.19 to 100.00]
  Role Functioning (C13, D1) (n=3, 3) | 88.90 [41.14 to 100.00] | 72.23 [9.00 to 100.00]
  Role Functioning (C14, D1) (n=2, 3) | 83.35 [0 to 100.00] | 66.67 [0 to 100.00]
  Role Functioning (C15, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | 83.35 [0 to 100.00]
  Role Functioning (C16, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | 66.65 [0 to 100.00]
  Role Functioning (C17, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | 58.35 [0 to 100.00]
  Role Functioning (C18, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | 66.65 [0 to 100.00]
  Cognitive Functioning (C1, D1) (n=49, 54) | 85.03 [78.76 to 91.31] | 82.71 [76.46 to 88.96]
  Cognitive Functioning (C2, D1) (n=41, 46) | 86.99 [81.16 to 92.81] | 82.24 [76.49 to 88.00]
  Cognitive Functioning (C3, D1) (n=27, 32) | 87.04 [77.13 to 96.94] | 82.29 [75.65 to 88.93]
  Cognitive Functioning (C4, D1) (n=19, 22) | 89.47 [80.91 to 98.03] | 81.06 [72.14 to 89.98]
  Cognitive Functioning (C5, D1) (n=14, 18) | 82.14 [64.65 to 99.62] | 81.48 [70.88 to 92.07]
  Cognitive Functioning (C6, D1) (n=8, 14) | 85.40 [76.47 to 94.33] | 84.53 [74.22 to 94.84]
  Cognitive Functioning (C7, D1) (n=7, 10) | 85.71 [71.86 to 99.57] | 89.99 [81.65 to 98.33]
  Cognitive Functioning (C8, D1) (n=4, 7) | 91.65 [76.31 to 100.00] | 71.43 [48.37 to 94.49]
  Cognitive Functioning (C9, D1) (n=4, 5) | 91.65 [76.31 to 100.00] | 83.34 [62.67 to 100.00]
  Cognitive Functioning (C10, D1) (n=3, 4) | 94.43 [70.48 to 100.00] | 79.18 [53.82 to 100.00]
  Cognitive Functioning (C11, D1) (n=3, 4) | 94.43 [70.48 to 100.00] | 87.50 [62.13 to 100.00]
  Cognitive Functioning (C12, D1) (n=3, 4) | 94.43 [70.48 to 100.00] | 79.15 [45.79 to 100.00]
  Cognitive Functioning (C13, D1) (n=3, 3) | 94.43 [70.48 to 100.00] | 83.33 [41.97 to 100.00]
  Cognitive Functioning (C14, D1) (n=2, 3) | 100.00 [100.00 to 100.00] | 83.33 [41.97 to 100.00]
  Cognitive Functioning (C15, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | 100.00 [100.00 to 100.00]
  Cognitive Functioning (C16, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | 91.65 [0 to 100.00]
  Cognitive Functioning (C17, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | 83.35 [0 to 100.00]
  Cognitive Functioning (C18, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | 100.00 [100.00 to 100.00]
  Emotional Functioning (C1, D1) (n=49, 53) | 74.65 [67.99 to 81.32] | 71.23 [64.54 to 77.92]
  Emotional Functioning (C2, D1) (n=41, 46) | 77.85 [71.07 to 84.62] | 71.37 [64.07 to 78.67]
  Emotional Functioning (C3, D1) (n=27, 32) | 76.86 [68.27 to 85.46] | 67.98 [58.91 to 77.04]
  Emotional Functioning (C4, D1) (n=19, 22) | 82.46 [76.06 to 88.87] | 71.21 [59.05 to 83.37]
  Emotional Functioning (C5, D1) (n=14, 18) | 79.18 [68.05 to 90.31] | 71.30 [58.02 to 84.58]
  Emotional Functioning (C6, D1) (n=8, 14) | 78.13 [62.35 to 93.90] | 79.76 [66.32 to 93.21]
  Emotional Functioning (C7, D1) (n=7, 10) | 79.77 [59.46 to 100.00] | 70.82 [53.89 to 87.75]
  Emotional Functioning (C8, D1) (n=4, 7) | 87.50 [62.13 to 100.00] | 61.90 [31.10 to 92.70]
  Emotional Functioning (C9, D1) (n=4, 5) | 91.68 [65.18 to 100.00] | 78.34 [47.67 to 100.00]
  Emotional Functioning (C10, D1) (n=3, 4) | 97.23 [85.33 to 100.00] | 66.68 [27.65 to 100.00]
  Emotional Functioning (C11, D1) (n=3, 4) | 97.23 [85.33 to 100.00] | 64.60 [23.56 to 100.00]
  Emotional Functioning (C12, D1) (n=3, 4) | 94.43 [70.48 to 100.00] | 54.15 [3.92 to 100.00]
  Emotional Functioning (C13, D1) (n=3, 3) | 86.13 [43.07 to 100.00] | 69.43 [0 to 100.00]
  Emotional Functioning (C14, D1) (n=2, 3) | 83.35 [0 to 100.00] | 63.90 [0 to 100.00]
  Emotional Functioning (C15, D1) (n=1, 2) | 91.70 [NA to NA] — number of participants in this category was 1 | 75.00 [0 to 100.00]
  Emotional Functioning (C16, D1) (n=1, 2) | 91.70 [NA to NA] — number of participants in this category was 1 | 75.00 [0 to 100.00]
  Emotional Functioning (C17, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | 62.50 [0 to 100.00]
  Emotional Functioning (C18, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | 83.35 [0 to 100.00]
  Social Functioning (C1, D1) (n=49, 53) | 80.95 [73.84 to 88.07] | 80.19 [72.98 to 87.40]
  Social Functioning (C2, D1) (n=41, 46) | 80.09 [72.26 to 87.91] | 77.53 [69.64 to 85.43]
  Social Functioning (C3, D1) (n=27, 32) | 79.01 [70.13 to 87.90] | 81.26 [73.67 to 88.85]
  Social Functioning (C4, D1) (n=19, 22) | 81.58 [73.60 to 89.56] | 75.75 [63.97 to 87.54]
  Social Functioning (C5, D1) (n=14, 18) | 76.19 [61.23 to 91.15] | 75.93 [64.48 to 87.37]
  Social Functioning (C6, D1) (n=8, 14) | 89.58 [79.21 to 99.94] | 80.96 [67.96 to 93.95]
  Social Functioning (C7, D1) (n=7, 10) | 90.47 [78.35 to 100.00] | 85.00 [74.57 to 95.43]
  Social Functioning (C8, D1) (n=4, 7) | 91.68 [65.18 to 100.00] | 73.81 [48.86 to 98.76]
  Social Functioning (C9, D1) (n=4, 5) | 91.68 [65.18 to 100.00] | 83.34 [62.67 to 100.00]
  Social Functioning (C10, D1) (n=3, 4) | 88.90 [41.14 to 100.00] | 83.33 [61.69 to 100.00]
  Social Functioning (C11, D1) (n=3, 4) | 94.43 [70.48 to 100.00] | 62.50 [0 to 100.00]
  Social Functioning (C12, D1) (n=3, 4) | 94.43 [70.48 to 100.00] | 66.68 [0 to 100.00]
  Social Functioning (C13, D1) (n=3, 3) | 88.90 [41.14 to 100.00] | 72.23 [0 to 100.00]
  Social Functioning (C14, D1) (n=2, 3) | 83.35 [0 to 100.00] | 72.20 [0 to 100.00]
  Social Functioning (C15, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | 91.65 [0 to 100.00]
  Social Functioning (C16, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | 91.65 [0 to 100.00]
  Social Functioning (C17, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | 83.35 [0 to 100.00]
  Social Functioning (C18, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | 91.65 [0 to 100.00]
  Fatigue (C1, D1) (n=49, 53) | 32.64 [25.95 to 39.33] | 33.11 [26.77 to 39.45]
  Fatigue (C2, D1) (n=41, 46) | 37.93 [30.24 to 45.62] | 39.85 [30.65 to 49.04]
  Fatigue (C3, D1) (n=28, 32) | 40.07 [30.81 to 49.34] | 37.49 [27.58 to 47.40]
  Fatigue (C4, D1) (n=19, 22) | 36.25 [23.77 to 48.74] | 33.84 [21.81 to 45.86]
  Fatigue (C5, D1) (n=14, 18) | 31.73 [18.69 to 44.77] | 44.44 [31.16 to 57.71]
  Fatigue (C6, D1) (n=9, 14) | 21.59 [11.04 to 32.13] | 33.32 [22.94 to 43.71]
  Fatigue (C7, D1) (n=7, 10) | 25.40 [3.41 to 47.39] | 33.32 [21.46 to 45.18]
  Fatigue (C8, D1) (n=4, 7) | 8.33 [0 to 25.24] | 39.69 [13.90 to 65.47]
  Fatigue (C9, D1) (n=4, 5) | 13.88 [0 to 40.37] | 28.90 [0 to 67.46]
  Fatigue (C10, D1) (n=3, 4) | 7.40 [0 to 39.24] | 36.10 [0 to 80.31]
  Fatigue (C11, D1) (n=3, 4) | 25.90 [0 to 83.30] | 30.55 [0 to 69.77]
  Fatigue (C12, D1) (n=3, 4) | 14.80 [0 to 78.48] | 27.78 [0 to 64.61]
  Fatigue (C13, D1) (n=3, 3) | 11.10 [0 to 58.86] | 25.90 [0 to 83.30]
  Fatigue (C14, D1) (n=2, 3) | 16.65 [0 to 100.00] | 40.73 [0 to 98.27]
  Fatigue (C15, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 100.00]
  Fatigue (C16, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 38.90 [0 to 100.00]
  Fatigue (C17, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 33.35 [0 to 100.00]
  Fatigue (C18, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 33.35 [0 to 100.00]
  Nausea/Vomiting (C1, D1) (n=49, 54) | 7.49 [3.33 to 11.64] | 9.26 [4.21 to 14.31]
  Nausea/Vomiting (C2, D1) (n=41, 46) | 16.26 [8.50 to 24.02] | 14.13 [7.62 to 20.65]
  Nausea/Vomiting (C3, D1) (n=28, 32) | 16.67 [6.87 to 26.46] | 11.98 [4.95 to 19.01]
  Nausea/Vomiting (C4, D1) (n=19, 22) | 13.16 [3.67 to 22.66] | 6.82 [1.40 to 12.24]
  Nausea/Vomiting (C5, D1) (n=14, 18) | 16.66 [0.21 to 33.11] | 8.34 [3.22 to 13.47]
  Nausea/Vomiting (C6, D1) (n=9, 14) | 9.26 [0 to 20.55] | 2.39 [0 to 5.89]
  Nausea/Vomiting (C7, D1) (n=7, 10) | 16.67 [0 to 40.22] | 8.34 [0 to 16.77]
  Nausea/Vomiting (C8, D1) (n=4, 7) | NA [NA to NA] — no participants reported this symptom at this time point | 9.51 [0 to 24.54]
  Nausea/Vomiting (C9, D1) (n=4, 5) | 4.18 [0 to 17.46] | 6.66 [0 to 25.15]
  Nausea/Vomiting (C10, D1) (n=3, 4) | 11.10 [0 to 58.86] | 12.50 [0 to 37.87]
  Nausea/Vomiting (C11, D1) (n=3, 4) | 16.67 [0 to 58.03] | 8.35 [0 to 23.69]
  Nausea/Vomiting (C12, D1) (n=3, 4) | 5.57 [0 to 29.52] | NA [NA to NA] — no participants reported this symptom at this time point
  Nausea/Vomiting (C17, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 8.35 [0 to 100.00]
  Pain (C1, D1) (n=49, 54) | 25.85 [18.67 to 33.04] | 30.25 [23.07 to 37.43]
  Pain (C2, D1) (n=41, 46) | 19.51 [11.21 to 27.82] | 31.52 [22.12 to 40.93]
  Pain (C3, D1) (n=28, 32) | 19.05 [10.48 to 27.61] | 28.65 [16.61 to 40.69]
  Pain (C4, D1) (n=19, 22) | 16.67 [6.30 to 27.04] | 28.80 [14.34 to 43.25]
  Pain (C5, D1) (n=14, 18) | 21.43 [3.96 to 38.90] | 33.34 [16.28 to 50.39]
  Pain (C6, D1) (n=9, 14) | 12.98 [0 to 29.66] | 25.00 [10.03 to 39.97]
  Pain (C7, D1) (n=7, 10) | 19.06 [0 to 41.63] | 23.34 [7.25 to 39.43]
  Pain (C8, D1) (n=4, 7) | 12.5 [0 to 37.87] | 19.04 [0.32 to 37.76]
  Pain (C9, D1) (n=4, 5) | 8.33 [0 to 34.82] | 20.00 [0 to 46.97]
  Pain (C10, D1) (n=3, 4) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 47.24]
  Pain (C11, D1) (n=3, 4) | NA [NA to NA] — no participants reported this symptom at this time point | 24.98 [0 to 51.47]
  Pain (C12, D1) (n=3, 4) | NA [NA to NA] — no participants reported this symptom at this time point | 24.98 [0 to 51.47]
  Pain (C13, D1) (n=3, 3) | 11.10 [0 to 58.86] | 22.20 [0 to 69.96]
  Pain (C14, D1) (n=2, 3) | 16.65 [0 to 100.00] | 22.20 [0 to 69.96]
  Pain (C16, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 100.00]
  Pain (C17, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 100.00]
  Pain (C18, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 100.00]
  Dyspnea (C1, D1) (n=49, 54) | 26.51 [20.04 to 32.99] | 25.91 [19.62 to 32.21]
  Dyspnea (C2, D1) (n=41, 46) | 30.07 [21.99 to 38.16] | 26.80 [19.39 to 34.21]
  Dyspnea (C3, D1) (n=28, 32) | 26.18 [15.42 to 36.94] | 24.99 [16.91 to 33.06]
  Dyspnea (C4, D1) (n=19, 22) | 36.83 [18.36 to 55.30] | 25.75 [12.90 to 38.60]
  Dyspnea (C5, D1) (n=14, 18) | 30.94 [13.29 to 48.59] | 29.62 [18.40 to 40.83]
  Dyspnea (C6, D1) (n=9, 14) | 25.91 [1.01 to 50.81] | 23.79 [14.77 to 32.80]
  Dyspnea (C7, D1) (n=7, 10) | 33.33 [8.14 to 58.51] | 19.98 [7.68 to 32.28]
  Dyspnea (C8, D1) (n=4, 7) | 16.65 [0 to 47.24] | 23.81 [0 to 53.15]
  Dyspnea (C9, D1) (n=4, 5) | 16.65 [0 to 47.24] | 6.66 [0 to 25.15]
  Dyspnea (C10, D1) (n=3, 4) | 22.23 [0 to 100.00] | 16.68 [0 to 69.74]
  Dyspnea (C11, D1) (n=3, 4) | 33.33 [0 to 100.00] | 8.33 [0 to 34.82]
  Dyspnea (C12, D1) (n=3, 4) | 22.23 [0 to 100.00] | 8.33 [0 to 34.82]
  Dyspnea (C13, D1) (n=3, 3) | 11.10 [0 to 58.86] | 22.20 [0 to 69.96]
  Dyspnea (C14, D1) (n=2, 3) | 16.65 [0 to 100.00] | 22.20 [0 to 69.96]
  Dyspnea (C15, D1) (n=1, 2) | 33.30 [NA to NA] — number of participants in this category was 1 | 16.65 [0 to 100.00]
  Dyspnea (C16, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 33.30 [33.30 to 33.30]
  Dyspnea (C17, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 33.35 [0 to 100.00]
  Dyspnea (C18, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 100.00]
  Insomnia (C1, D1) (n=49, 54) | 29.24 [19.74 to 38.75] | 27.78 [18.30 to 37.26]
  Insomnia (C2, D1) (n=41, 46) | 22.76 [12.66 to 32.86] | 29.71 [19.87 to 39.55]
  Insomnia (C3, D1) (n=28, 32) | 29.75 [17.91 to 41.60] | 38.54 [25.19 to 51.89]
  Insomnia (C4, D1) (n=19, 22) | 14.03 [4.28 to 23.78] | 25.76 [11.38 to 40.14]
  Insomnia (C5, D1) (n=14, 18) | 19.04 [2.65 to 35.42] | 33.33 [18.28 to 48.37]
  Insomnia (C6, D1) (n=9, 14) | 11.10 [0 to 23.90] | 23.81 [7.92 to 39.70]
  Insomnia (C7, D1) (n=7, 10) | 14.29 [0 to 38.55] | 19.99 [3.32 to 36.66]
  Insomnia (C8, D1) (n=4, 7) | 33.33 [0 to 76.65] | 38.09 [5.12 to 71.05]
  Insomnia (C9, D1) (n=4, 5) | 24.98 [0 to 51.47] | 33.32 [0 to 84.01]
  Insomnia (C10, D1) (n=3, 4) | 22.23 [0 to 100.00] | 41.68 [0 to 92.49]
  Insomnia (C11, D1) (n=3, 4) | 33.33 [0 to 100.00] | 33.33 [0 to 76.65]
  Insomnia (C12, D1) (n=3, 4) | 33.33 [0 to 100.00] | 16.65 [0 to 47.24]
  Insomnia (C13, D1) (n=3, 3) | 22.20 [0 to 69.96] | 22.20 [0 to 69.96]
  Insomnia (C14, D1) (n=2, 3) | 33.30 [33.30 to 33.30] | 44.47 [0 to 100.00]
  Insomnia (C15, D1) (n=1, 2) | 33.30 [NA to NA] — number of participants in this category was 1 | 16.65 [0 to 100.00]
  Insomnia (C16, D1) (n=1, 2) | 33.30 [NA to NA] — number of participants in this category was 1 | 16.65 [0 to 100.00]
  Insomnia (C17, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 100.00]
  Insomnia (C18, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 100.00]
  Loss of Appetite (C1, D1) (n=49, 54) | 23.12 [14.78 to 31.46] | 20.99 [13.42 to 28.55]
  Loss of Appetite (C2, D1) (n=41, 46) | 33.33 [22.04 to 44.61] | 26.81 [17.56 to 36.05]
  Loss of Appetite (C3, D1) (n=28, 32) | 36.90 [22.68 to 51.12] | 26.04 [14.32 to 37.76]
  Loss of Appetite (C4, D1) (n=19, 22) | 28.06 [11.76 to 44.36] | 24.24 [8.99 to 39.49]
  Loss of Appetite (C5, D1) (n=14, 18) | 26.18 [12.72 to 39.64] | 24.08 [7.20 to 40.95]
  Loss of Appetite (C6, D1) (n=9, 14) | 22.21 [4.09 to 40.33] | 26.19 [5.96 to 46.42]
  Loss of Appetite (C7, D1) (n=7, 10) | 28.56 [7.28 to 49.83] | 30.00 [0 to 60.68]
  Loss of Appetite (C8, D1) (n=4, 7) | 16.65 [0 to 47.24] | 14.29 [0 to 38.55]
  Loss of Appetite (C9, D1) (n=4, 5) | 16.65 [0 to 47.24] | 20.00 [0 to 57.03]
  Loss of Appetite (C10, D1) (n=3, 4) | 22.23 [0 to 100.00] | 25.00 [0 to 75.80]
  Loss of Appetite (C11, D1) (n=3, 4) | 22.23 [0 to 100.00] | 33.33 [0 to 100.00]
  Loss of Appetite (C12, D1) (n=3, 4) | 22.20 [0 to 69.96] | 25.00 [0 to 75.80]
  Loss of Appetite (C13, D1) (n=3, 3) | 22.20 [0 to 69.96] | 11.10 [0 to 58.86]
  Loss of Appetite (C14, D1) (n=2, 3) | 16.65 [0 to 100.00] | 11.10 [0 to 58.86]
  Loss of Appetite (C17, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 100.00]
  Constipation (C1, D1) (n=48, 54) | 12.49 [6.63 to 18.36] | 16.67 [9.65 to 23.68]
  Constipation (C2, D1) (n=41, 46) | 4.88 [0 to 9.90] | 13.77 [5.53 to 22.00]
  Constipation (C3, D1) (n=28, 32) | 13.10 [2.34 to 23.85] | 18.75 [6.56 to 30.94]
  Constipation (C4, D1) (n=19, 22) | 1.75 [0 to 5.43] | 10.60 [0.02 to 21.18]
  Constipation (C5, D1) (n=14, 18) | 7.14 [0 to 15.32] | 14.82 [1.82 to 27.81]
  Constipation (C6, D1) (n=8, 13) | 12.50 [0 to 33.24] | 12.82 [0 to 25.92]
  Constipation (C7, D1) (n=7, 10) | 4.76 [0 to 16.40] | 3.33 [0 to 10.86]
  Constipation (C8, D1) (n=4, 7) | 8.33 [0 to 34.82] | NA [NA to NA] — no participants reported this symptom at this time point
  Constipation (C9, D1) (n=4, 5) | 8.33 [0 to 34.82] | 13.34 [0 to 50.38]
  Constipation (C10, D1) (n=3, 4) | NA [NA to NA] — no participants reported this symptom at this time point | 8.33 [0 to 34.82]
  Constipation (C11, D1) (n=3, 4) | NA [NA to NA] — no participants reported this symptom at this time point | 8.33 [0 to 34.82]
  Constipation (C12, D1) (n=3, 4) | 11.10 [0 to 58.86] | 8.33 [0 to 34.82]
  Constipation (C13, D1) (n=3, 3) | 11.10 [0 to 58.86] | NA [NA to NA] — no participants reported this symptom at this time point
  Constipation (C14, D1) (n=2, 3) | 16.65 [0 to 100.00] | NA [NA to NA] — no participants reported this symptom at this time point
  Constipation (C15, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 100]
  Diarrhea (C1, D1) (n=49, 54) | 6.80 [2.02 to 11.58] | 2.47 [0.06 to 4.87]
  Diarrhea (C2, D1) (n=41, 46) | 38.21 [28.35 to 48.07] | 21.01 [13.97 to 28.04]
  Diarrhea (C3, D1) (n=27, 32) | 37.03 [23.68 to 50.39] | 17.69 [9.63 to 25.76]
  Diarrhea (C4, D1) (n=19, 22) | 38.59 [23.19 to 53.99] | 7.57 [1.24 to 13.90]
  Diarrhea (C5, D1) (n=14, 18) | 30.94 [16.89 to 45.00] | 14.81 [4.60 to 25.01]
  Diarrhea (C6, D1) (n=8, 14) | 24.99 [5.28 to 44.69] | 11.90 [0 to 24.09]
  Diarrhea (C7, D1) (n=7, 10) | 42.86 [19.53 to 66.18] | 6.66 [0 to 16.70]
  Diarrhea (C8, D1) (n=4, 7) | 33.30 [33.30 to 33.30] | 14.29 [0 to 38.55]
  Diarrhea (C9, D1) (n=4, 5) | 33.30 [33.30 to 33.30] | 6.66 [0 to 25.15]
  Diarrhea (C10, D1) (n=3, 4) | 33.33 [0 to 100.00] | 8.33 [0 to 34.82]
  Diarrhea (C11, D1) (n=3, 4) | 33.33 [0 to 100.00] | 16.65 [0 to 47.24]
  Diarrhea (C12, D1) (n=3, 4) | 66.67 [0 to 100.00] | 16.65 [0 to 47.24]
  Diarrhea (C13, D1) (n=3, 3) | 33.30 [33.30 to 33.30] | 11.10 [0 to 58.86]
  Diarrhea (C14, D1) (n=2, 3) | 50.00 [0 to 100.00] | 11.10 [0 to 58.86]
  Diarrhea (C15, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 100.00]
  Diarrhea (C16, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 100.00]
  Diarrhea (C17, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 100.00]
  Diarrhea (C18, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 100.00]
  Financial Difficulties (C1, D1) (n=49, 53) | 21.76 [12.69 to 30.84] | 13.84 [6.31 to 21.36]
  Financial Difficulties (C2, D1) (n=41, 45) | 17.07 [8.88 to 25.26] | 11.85 [4.40 to 19.29]
  Financial Difficulties (C3, D1) (n=27, 32) | 17.27 [8.80 to 25.75] | 16.66 [7.01 to 26.32]
  Financial Difficulties (C4, D1) (n=19, 22) | 8.77 [0 to 17.80] | 24.25 [8.32 to 40.17]
  Financial Difficulties (C5, D1) (n=14, 18) | 21.42 [3.55 to 39.30] | 16.67 [2.45 to 30.89]
  Financial Difficulties (C6, D1) (n=8, 14) | 24.99 [5.28 to 44.69] | 19.05 [0 to 38.61]
  Financial Difficulties (C7, D1) (n=7, 10) | 9.51 [0 to 24.54] | 13.33 [0 to 36.37]
  Financial Difficulties (C8, D1) (n=4, 7) | 41.65 [0 to 100.00] | 38.10 [0 to 83.23]
  Financial Difficulties (C9, D1) (n=4, 5) | 33.33 [0 to 100.00] | 26.66 [0 to 80.62]
  Financial Difficulties (C10, D1) (n=3, 4) | 44.43 [0 to 100.00] | 33.33 [0 to 100.00]
  Financial Difficulties (C11, D1) (n=3, 4) | 44.43 [0 to 100.00] | 33.33 [0 to 100.00]
  Financial Difficulties (C12, D1) (n=3, 4) | 44.43 [0 to 100.00] | 33.33 [0 to 100.00]
  Financial Difficulties (C13, D1) (n=3, 3) | 44.43 [0 to 100.00] | 33.33 [0 to 100.00]
  Financial Difficulties (C14, D1) (n=2, 3) | 66.65 [0 to 100.00] | 33.33 [0 to 100.00]
  Financial Difficulties (C15, D1) (n=1, 2) | 100.00 [NA to NA] — number of participants in this category was 1 | NA [NA to NA] — no participants reported this symptom at this time point
  Financial Difficulties (C16, D1) (n=1, 2) | 100 [NA to NA] — number of participants in this category was 1 | NA [NA to NA] — no participants reported this symptom at this time point

59. Other Pre Specified Outcome: sKIT Ratio to Baseline at Each Timepoint
Description: Plasma sKIT concentration at each time point divided by sKIT concentration at baseline (ratio to baseline)
Time Frame: Baseline to Cycle 2 (Day 1) and Cycle 3 (Day 1)
Population: FA Set; n equals number of participants with evaluable data at specified cycle
Measure: Median (Full Range); unit: Ratio
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
Ratio
  Cycle 2, Day 1 (n=43, 47) | 0.76 [0.38 to 1.33] | 1.00 [0.61 to 1.44]
  Cycle 3, Day 1 (n=36, 36) | 0.58 [0.22 to 1.05] | 0.95 [0.45 to 1.51]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; sKIT Ratio to Baseline for Cycle 2, Day 1; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; sKIT Ratio to Baseline for Cycle 3, Day 1; Test type: Superiority or Other; p < 0.0001, Wilcoxon Rank Sum Test

60. Secondary Outcome: EORTC-QLQ-C30 Lung Cancer Module (LC13) Score
Description: The EORTC-QLQ-C30 LC13 is a self-administered questionnaire assessing specific lung cancer disease related symptoms (dyspnea, coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, pain in the chest, arm/shoulder or other parts of the body). Recall period: past week; response range: not at all (1) to very much (4). Scale score range: 0 to 100. Higher symptom score = greater degree of symptoms.
Time Frame: Baseline (Cycle 1 [Day 1]) to Cycle 18 (Day 1)
Population: PRO Analysis Set; n is number of participants with an assessment at the specific time point
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 49 | 54
score on a scale
  Dyspnea Symptom (C1, D1) (n=48, 53) | 21.05 [15.64 to 26.47] | 25.56 [19.57 to 31.56]
  Dyspnea Symptom (C2, D1) (n=38, 46) | 25.71 [20.33 to 31.09] | 26.08 [19.04 to 33.11]
  Dyspnea Symptom (C3, D1) (n=26, 32) | 24.77 [17.02 to 32.52] | 26.03 [18.31 to 33.76]
  Dyspnea Symptom (C4, D1) (n=18, 22) | 27.16 [13.85 to 40.46] | 23.73 [13.84 to 33.61]
  Dyspnea Symptom (C5, D1) (n=12, 18) | 22.21 [9.44 to 34.98] | 32.71 [22.07 to 43.35]
  Dyspnea Symptom (C6, D1) (n=8, 14) | 18.04 [7.02 to 29.06] | 21.41 [11.85 to 30.97]
  Dyspnea Symptom (C7, D1) (n=6, 10) | 14.80 [0.69 to 28.91] | 29.99 [18.70 to 41.28]
  Dyspnea Symptom (C8, D1) (n=4, 6) | 8.33 [0 to 25.24] | 22.22 [0 to 46.68]
  Dyspnea Symptom (C9, D1) (n=4, 3) | 11.10 [0 to 31.49] | 22.20 [0 to 77.35]
  Dyspnea Symptom (C10, D1) (n=3, 4) | 11.10 [0 to 58.86] | 33.33 [0 to 78.99]
  Dyspnea Symptom (C11, D1) (n=3, 3) | 18.50 [0 to 60.62] | 29.60 [0 to 93.28]
  Dyspnea Symptom (C12, D1) (n=3, 4) | 14.80 [0 to 78.48] | 22.20 [0 to 47.18]
  Dyspnea Symptom (C13, D1) (n=3, 3) | 7.40 [0 to 39.24] | 22.20 [0 to 77.35]
  Dyspnea Symptom (C14, D1) (n=2, 3) | 16.65 [0 to 87.17] | 25.90 [0 to 83.30]
  Dyspnea Symptom (C15, D1) (n=1, 2) | 22.20 [NA to NA] — number of participants in this category was 1 | 11.10 [0 to 100.00]
  Dyspnea Symptom (C16, D1) (n=1, 2) | NA [NA to NA] — number of participants in this category was 1 | 22.20 [0 to 100.00]
  Dyspnea Symptom (C17, D1) (n=1, 2) | NA [NA to NA] — number of participants in this category was 1 | 22.20 [0 to 100.00]
  Dyspnea Symptom (C18, D1) (n=1, 2) | NA [NA to NA] — number of participants in this category was 1 | 16.65 [0 to 100.00]
  Coughing Symptom (C1, D1) (n=49, 53) | 36.72 [29.09 to 44.36] | 37.10 [29.31 to 44.88]
  Coughing Symptom (C2, D1) (n=41, 46) | 31.70 [22.91 to 40.49] | 31.87 [24.65 to 39.09]
  Coughing Symptom (C3, D1) (n=27, 32) | 32.09 [20.82 to 43.35] | 30.20 [19.04 to 41.36]
  Coughing Symptom (C4, D1) (n=19, 22) | 29.81 [16.81 to 42.81] | 15.14 [7.61 to 22.66]
  Coughing Symptom (C5, D1) (n=14, 18) | 38.08 [23.25 to 52.91] | 29.62 [17.05 to 42.20]
  Coughing Symptom (C6, D1) (n=9, 14) | 33.31 [11.12 to 55.50] | 26.17 [15.03 to 37.31]
  Coughing Symptom (C7, D1) (n=7, 10) | 33.33 [8.14 to 58.51] | 16.67 [0 to 36.94]
  Coughing Symptom (C8, D1) (n=4, 7) | 24.98 [0 to 51.47] | 28.56 [7.28 to 49.83]
  Coughing Symptom (C9, D1) (n=4, 4) | 24.98 [0 to 51.47] | 8.33 [0 to 34.82]
  Coughing Symptom (C10, D1) (n=3, 4) | 22.20 [0 to 69.96] | 25.00 [0 to 75.80]
  Coughing Symptom (C11, D1) (n=3, 3) | 22.20 [0 to 69.96] | 33.33 [0 to 100.00]
  Coughing Symptom (C12, D1) (n=3, 4) | 22.20 [0 to 69.96] | 41.65 [15.08 to 68.22]
  Coughing Symptom (C13, D1) (n=3, 3) | 22.20 [0 to 69.96] | 33.33 [0 to 100.00]
  Coughing Symptom (C14, D1) (n=2, 3) | 16.65 [0 to 100.00] | 11.10 [0 to 58.86]
  Coughing Symptom (C15, D1) (n=1, 2) | NA [NA to NA] — number of participants in this category was 1 | 16.65 [0 to 100.00]
  Coughing Symptom (C16, D1) (n=1, 2) | NA [NA to NA] — number of participants in this category was 1 | 16.65 [0 to 100.00]
  Coughing Symptom (C17, D1) (n=1, 2) | NA [NA to NA] — number of participants in this category was 1 | 16.65 [0 to 100.00]
  Coughing Symptom (C18, D1) (n=1, 2) | NA [NA to NA] — number of participants in this category was 1 | 33.35 [0 to 100.00]
  Haemoptysis Symptom (C1, D1) (n=49, 54) | 2.04 [0 to 4.36] | 6.17 [0.85 to 11.50]
  Haemoptysis Symptom (C2, D1) (n=41, 46) | 6.50 [0.18 to 12.82] | 4.34 [0.98 to 7.71]
  Haemoptysis Symptom (C3, D1) (n=27, 32) | 2.47 [0 to 5.98] | 5.21 [0 to 10.59]
  Haemoptysis Symptom (C4, D1) (n=19, 22) | 1.75 [0 to 5.43] | 1.51 [0 to 4.66]
  Haemoptysis Symptom (C5, D1) (n=14, 18) | 2.38 [0 to 7.52] | 5.56 [0 to 14.09]
  Haemoptysis Symptom (C6, D1) (n=9, 14) | 3.70 [0 to 12.23] | 2.38 [0 to 7.52]
  Haemoptysis Symptom (C7, D1) (n=7, 10) | 4.76 [0 to 16.40] | NA [NA to NA] — no participants reported this symptom at this time point
  Haemoptysis Symptom (C8, D1) (n=4, 6) | NA [NA to NA] — no participants reported this symptom at this time point | 5.55 [0 to 19.82]
  Sore Mouth Symptom (C1, D1) (n=49, 54) | 6.12 [1.90 to 10.34] | 1.23 [0 to 2.97]
  Sore Mouth Symptom (C2, D1) (n=41, 46) | 19.50 [11.36 to 27.65] | 7.97 [3.22 to 12.71]
  Sore Mouth Symptom (C3, D1) (n=27, 32) | 16.04 [6.11 to 25.97] | 6.25 [0 to 12.68]
  Sore Mouth Symptom (C4, D1) (n=19, 22) | 12.27 [0.05 to 24.50] | 7.58 [0 to 16.62]
  Sore Mouth Symptom (C5, D1) (n=14, 18) | 23.79 [7.91 to 39.68] | 12.96 [0 to 27.05]
  Sore Mouth Symptom (C6, D1) (n=9, 14) | 11.10 [0 to 23.90] | 2.38 [0 to 7.52]
  Sore Mouth Symptom (C7, D1) (n=7, 10) | 4.76 [0 to 16.40] | 6.67 [0 to 21.76]
  Sore Mouth Symptom (C8, D1) (n=4, 6) | NA [NA to NA] — no participants reported this symptom at this time point | 5.55 [0 to 19.82]
  Sore Mouth Symptom (C10, D1) (n=3, 4) | NA [NA to NA] — no participants reported this symptom at this time point | 8.33 [0 to 34.82]
  Sore Mouth Symptom (C13, D1) (n=3, 3) | NA [NA to NA] — no participants reported this symptom at this time point | 11.10 [0 to 58.86]
  Sore Mouth Symptom (C14, D1) (n=2, 3) | NA [NA to NA] — no participants reported this symptom at this time point | 11.10 [0 to 58.86]
  Dysphagia Symptom (C1, D1) (n=49, 54) | 6.80 [2.02 to 11.58] | 6.17 [1.47 to 10.87]
  Dysphagia Symptom (C2, D1) (n=41, 46) | 13.00 [5.99 to 20.01] | 10.14 [3.93 to 16.35]
  Dysphagia Symptom (C3, D1) (n=26, 32) | 7.68 [1.91 to 13.46] | 14.58 [3.19 to 25.98]
  Dysphagia Symptom (C4, D1) (n=19, 22) | 7.01 [0.29 to 13.73] | 12.12 [0.45 to 23.79]
  Dysphagia Symptom (C5, D1) (n=14, 18) | 11.91 [0 to 26.25] | 11.11 [0 to 25.04]
  Dysphagia Symptom (C6, D1) (n=9, 14) | 3.70 [0 to 12.23] | 7.14 [0 to 15.32]
  Dysphagia Symptom (C7, D1) (n=7, 10) | 4.76 [0 to 16.40] | 10.00 [0 to 26.10]
  Dysphagia Symptom (C8, D1) (n=4, 6) | 8.33 [0 to 34.82] | NA [NA to NA] — no participants reported this symptom at this time point
  Dysphagia Symptom (C9, D1) (n=4, 3) | 8.33 [0 to 34.82] | NA [NA to NA] — no participants reported this symptom at this time point
  Dysphagia Symptom (C10, D1) (n=3, 4) | 22.23 [0 to 100.00] | 16.65 [0 to 47.24]
  Dysphagia Symptom (C11, D1) (n=3, 3) | 11.10 [0 to 58.86] | NA [NA to NA] — no participants reported this symptom at this time point
  Dysphagia Symptom (C12, D1) (n=3, 4) | 22.23 [0 to 100.0] | 8.33 [0 to 34.82]
  Dysphagia Symptom (C13, D1) (n=3, 3) | NA [NA to NA] — no participants reported this symptom at this time point | 22.20 [0 to 69.96]
  Dysphagia Symptom (C14, D1) (n=2, 3) | NA [NA to NA] — no participants reported this symptom at this time point | 11.10 [0 to 58.86]
  Peripheral Neuropathy Symptom (C1, D1) (n=49, 54) | 18.37 [9.83 to 26.90] | 17.28 [9.42 to 25.13]
  Peripheral Neuropathy Symptom (C2, D1) (n=41, 46) | 14.63 [7.17 to 22.09] | 20.28 [11.81 to 28.75]
  Peripheral Neuropathy Symptom (C3, D1) (n=27, 32) | 16.04 [5.46 to 26.63] | 34.37 [19.89 to 48.84]
  Peripheral Neuropathy Symptom (C4, D1) (n=19, 22) | 22.81 [7.61 to 38.00] | 25.75 [12.12 to 39.39]
  Peripheral Neuropathy Symptom (C5, D1) (n=14, 18) | 26.18 [12.72 to 39.64] | 22.22 [8.29 to 36.15]
  Peripheral Neuropathy Symptom (C6, D1) (n=9, 14) | 18.51 [0 to 37.13] | 23.81 [7.92 to 39.70]
  Peripheral Neuropathy Symptom (C7, D1) (n=7, 10) | 33.33 [8.14 to 58.51] | 23.33 [3.69 to 42.97]
  Peripheral Neuropathy Symptom (C8, D1) (n=4, 6) | 24.98 [0 to 51.47] | 22.20 [4.15 to 40.25]
  Peripheral Neuropathy Symptom (C9, D1) (n=4, 3) | 16.65 [0 to 47.24] | 33.30 [33.30 to 33.30]
  Peripheral Neuropathy Symptom (C10, D1) (n=3, 4) | NA [NA to NA] — no participants reported this symptom at this time point | 33.30 [33.30 to 33.30]
  Peripheral Neuropathy Symptom (C11, D1) (n=3, 3) | 22.20 [0 to 69.96] | 44.43 [0 to 92.34]
  Peripheral Neuropathy Symptom (C12, D1) (n=3, 4) | 22.23 [0 to 100.00] | 41.65 [15.08 to 68.22]
  Peripheral Neuropathy Symptom (C13, D1) (n=3, 3) | 11.10 [0 to 58.86] | 44.43 [0 to 92.34]
  Peripheral Neuropathy Symptom (C14, D1) (n=2, 3) | 16.65 [0 to 100.00] | 44.43 [0 to 92.34]
  Peripheral Neuropathy Symptom (C15, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 100.00]
  Peripheral Neuropathy Symptom (C16, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 100.00]
  Peripheral Neuropathy Symptom (C17, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 33.30 [33.30 to 33.30]
  Peripheral Neuropathy Symptom (C18, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 33.30 [33.30 to 33.30]
  Alopecia Symptom (C1, D1) (n=49, 54) | 12.92 [5.40 to 20.45] | 12.96 [4.98 to 20.95]
  Alopecia Symptom (C2, D1) (n=41, 46) | 4.87 [1.11 to 8.63] | 5.79 [1.47 to 10.12]
  Alopecia Symptom (C3, D1) (n=27, 32) | 7.40 [0.73 to 14.08] | 5.20 [0.77 to 9.63]
  Alopecia Symptom (C4, D1) (n=19, 22) | 10.52 [0 to 22.56] | 13.63 [1.86 to 25.40]
  Alopecia Symptom (C5, D1) (n=14, 18) | 16.66 [4.14 to 29.17] | 22.22 [9.50 to 34.93]
  Alopecia Symptom (C6, D1) (n=9, 14) | 14.80 [1.31 to 28.29] | 19.04 [2.65 to 35.42]
  Alopecia Symptom (C7, D1) (n=7, 10) | 14.27 [0 to 30.73] | 16.67 [0 to 36.94]
  Alopecia Symptom (C8, D1) (n=4, 6) | 8.33 [0 to 34.82] | 11.10 [0 to 29.15]
  Alopecia Symptom (C9, D1) (n=4, 3) | 16.65 [0 to 47.24] | 22.23 [0 to 100.00]
  Alopecia Symptom (C10, D1) (n=3, 4) | 11.10 [0 to 58.86] | 25.00 [0 to 75.80]
  Alopecia Symptom (C11, D1) (n=3, 3) | 33.30 [33.30 to 33.30] | NA [NA to NA] — no participants reported this symptom at this time point
  Alopecia Symptom (C12, D1) (n=3, 4) | 33.33 [0 to 100.00] | 25.00 [0 to 75.80]
  Alopecia Symptom (C13, D1) (n=3, 3) | 33.30 [33.30 to 33.30] | 33.33 [0 to 100.00]
  Alopecia Symptom (C14, D1) (n=2, 3) | 33.35 [0 to 100.00] | 33.33 [0 to 100.00]
  Pain in Chest Symptom (C1, D1) (n=49, 53) | 19.72 [11.93 to 27.52] | 15.09 [8.70 to 21.47]
  Pain in Chest Symptom (C2, D1) (n=41, 46) | 11.38 [4.48 to 18.28] | 14.48 [6.50 to 22.47]
  Pain in Chest Symptom (C3, D1) (n=27, 32) | 8.64 [1.71 to 15.57] | 18.75 [8.65 to 28.84]
  Pain in Chest Symptom (C4, D1) (n=18, 22) | 11.11 [1.26 to 20.95] | 10.60 [0 to 22.13]
  Pain in Chest Symptom (C5, D1) (n=14, 18) | 16.66 [0.21 to 33.11] | 20.37 [4.15 to 36.60]
  Pain in Chest Symptom (C6, D1) (n=9, 14) | 11.10 [0 to 23.90] | 11.90 [0 to 24.09]
  Pain in Chest Symptom (C7, D1) (n=7, 10) | 19.03 [2.57 to 35.49] | 16.66 [0 to 39.83]
  Pain in Chest Symptom (C8, D1) (n=4, 6) | 8.33 [0 to 34.82] | 5.55 [0 to 19.82]
  Pain in Chest Symptom (C9, D1) (n=4, 3) | 8.33 [0 to 34.82] | NA [NA to NA] — no participants reported this symptom at this time point
  Pain in Chest Symptom (C10, D1) (n=3, 4) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 47.24]
  Pain in Chest Symptom (C11, D1) (n=3, 3) | NA [NA to NA] — no participants reported this symptom at this time point | 11.10 [0 to 58.86]
  Pain in Chest Symptom (C12, D1) (n=3, 4) | NA [NA to NA] — no participants reported this symptom at this time point | 8.33 [0 to 34.82]
  Pain in Chest Symptom (C13, D1) (n=3, 3) | 11.10 [0 to 58.86] | 22.20 [0 to 69.96]
  Pain in Chest Symptom (C14, D1) (n=2, 3) | 16.65 [0 to 100.00] | 11.10 [0 to 58.86]
  Pain in Chest Symptom (C16, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 100.00]
  Pain in Chest Symptom (C17, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 100.00]
  Pain in Arm or Shoulder (C1, D1) (n=49, 54) | 21.08 [14.12 to 28.05] | 11.72 [6.09 to 17.36]
  Pain in Arm or Shoulder (C2, D1) (n=41, 46) | 10.56 [5.08 to 16.04] | 16.66 [9.82 to 23.50]
  Pain in Arm or Shoulder (C3, D1) (n=27, 32) | 14.81 [6.36 to 23.25] | 17.71 [7.59 to 27.82]
  Pain in Arm or Shoulder (C4, D1) (n=19, 22) | 12.27 [4.31 to 20.22] | 21.21 [7.87 to 34.54]
  Pain in Arm or Shoulder (C5, D1) (n=14, 18) | 19.04 [2.65 to 35.42] | 25.92 [10.29 to 41.55]
  Pain in Arm or Shoulder (C6, D1) (n=9, 14) | 14.80 [1.31 to 28.29] | 26.19 [7.42 to 44.95]
  Pain in Arm or Shoulder (C7, D1) (n=7, 10) | 23.80 [0.49 to 47.11] | 23.33 [0 to 48.59]
  Pain in Arm or Shoulder (C8, D1) (n=4, 6) | 16.65 [0 to 47.24] | 5.55 [0 to 19.82]
  Pain in Arm or Shoulder (C9, D1) (n=4, 3) | 16.65 [0 to 47.24] | 11.10 [0 to 58.86]
  Pain in Arm or Shoulder (C10, D1) (n=3, 4) | 11.10 [0 to 58.86] | 8.33 [0 to 34.82]
  Pain in Arm or Shoulder (C11, D1) (n=3, 3) | 11.10 [0 to 58.86] | 11.10 [0 to 58.86]
  Pain in Arm or Shoulder (C12, D1) (n=3, 4) | 11.10 [0 to 58.86] | 8.33 [0 to 34.82]
  Pain in Arm or Shoulder (C13, D1) (n=3, 3) | 22.20 [0 to 69.96] | 22.20 [0 to 69.96]
  Pain in Arm or Shoulder (C14, D1) (n=2, 3) | 16.65 [0 to 100.00] | 11.10 [0 to 58.86]
  Pain in Arm or Shoulder (C15, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 100.00]
  Pain in Arm or Shoulder (C16, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 100.00]
  Pain in Arm or Shoulder (C17, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 100.00]
  Pain in Arm or Shoulder (C18, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 100.00]
  Pain in Other Parts of Body (C1, D1) (n=48, 51) | 26.38 [16.61 to 36.16] | 35.29 [26.61 to 43.97]
  Pain in Other Parts of Body (C2, D1) (n=40, 43) | 14.17 [6.57 to 21.76] | 28.68 [18.04 to 39.32]
  Pain in Other Parts of Body (C3, D1) (n=26, 31) | 16.67 [6.41 to 26.92] | 29.03 [15.73 to 42.33]
  Pain in Other Parts of Body (C4, D1) (n=18, 20) | 14.81 [0.63 to 28.99] | 20.00 [6.23 to 33.76]
  Pain in Other Parts of Body (C5, D1) (n=13, 18) | 35.90 [11.98 to 59.82] | 31.48 [13.98 to 48.98]
  Pain in Other Parts of Body (C6, D1) (n=9, 14) | 18.51 [0 to 37.13] | 21.43 [5.22 to 37.64]
  Pain in Other Parts of Body (C7, D1) (n=6, 10) | 16.67 [0 to 45.94] | 33.34 [5.80 to 60.88]
  Pain in Other Parts of Body (C8, D1) (n=4, 6) | NA [NA to NA] — no participants reported this symptom at this time point | 27.77 [1.43 to 54.11]
  Pain in Other Parts of Body (C9, D1) (n=4, 3) | NA [NA to NA] — no participants reported this symptom at this time point | 22.20 [0 to 69.96]
  Pain in Other Parts of Body (C10, D1) (n=3, 4) | NA [NA to NA] — no participants reported this symptom at this time point | 8.33 [0 to 34.82]
  Pain in Other Parts of Body (C11, D1) (n=3, 3) | NA [NA to NA] — no participants reported this symptom at this time point | 11.10 [0 to 58.86]
  Pain in Other Parts of Body (C12, D1) (n=3, 4) | NA [NA to NA] — no participants reported this symptom at this time point | 8.33 [0 to 34.82]
  Pain in Other Parts of Body (C13, D1) (n=3, 3) | NA [NA to NA] — no participants reported this symptom at this time point | 22.20 [0 to 69.96]
  Pain in Other Parts of Body (C14, D1) (n=2, 3) | 16.65 [0 to 100.00] | NA [NA to NA] — no participants reported this symptom at this time point
  Pain in Other Parts of Body (C16, D1) (n=1, 2) | NA [NA to NA] — no participants reported this symptom at this time point | 16.65 [0 to 100.00]

61. Secondary Outcome: Number of Participants With Blood Pressure (BP) Greater Than 150/100 Millimeters of Mercury (mmHg)
Description: Systolic/diastolic BP measured in triplicate (separated by approximately 2 minutes [min]) using validated electronic device (same device for all measurements), recorded to nearest mmHg. Dominant arm used (same one each time) with appropriate cuff size encircling at least 80% of arm. BP measured after 5 min rest and before invasive procedures, while seated in a chair with back supported, arms bared, supported at heart level. No smoking or caffeine use allowed during 30 min before measurement. Number of participants with systolic BP >150 mmHg/diastolic BP >100 mmHg at any timepoint postbaseline.
Time Frame: Randomization up until Month 17
Population: Per-Protocol Set: all participants in the Phase 2 portion (randomized) who received at least 1 dose of study medication (either erlotinib or blinded medication) with treatment assignments designated according to actual study medication received
Measure: Number; unit: Participants
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 64 | 64
Participants | 10 | 8

62. Secondary Outcome: Number of Participants With BP Greater Than 200/110 mmHg
Description: as for outcome 61
Time Frame: Randomization up until Month 17
Population: Per-Protocol Set
Measure: Number; unit: Participants
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 64 | 64
Participants | 1 | 0

63. Secondary Outcome: Number of Participants on Anti-hypertensive Medications
Description: Number of participants with BP greater than 150/100 mmHg or 200/110 mmHg who were treated with anti-hypertensive medications.
Time Frame: Randomization to Day 28 of Cycle 18
Population: Per Protocol Set; data were not analyzed
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 0 | 0

64. Secondary Outcome: Plasma Concentration of VEGF-C at Baseline
Time Frame: Baseline (Cycle 1, Day 1)
Population: FA Set
Measure: Median (Full Range); unit: picograms (pg)/mL
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
picograms (pg)/mL | 474.15 [190.40 to 2469.80] | 502.10 [255.50 to 1921.50]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Test type: Superiority or Other; p = 0.3681, Wilcoxon Rank Sum Test — 2-sided normal approximated p-value

65. Secondary Outcome: Plasma Concentration of Soluble VEGFR-2 at Baseline
Time Frame: Baseline (Cycle 1, Day 1)
Population: FA Set
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
pg/mL | 10904.50 [6320 to 17733] | 10027 [7592.50 to 18363]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Test type: Superiority or Other; p = 0.5982, Wilcoxon Rank Sum Test — 2-sided normal approximated p-value

66. Secondary Outcome: Plasma Concentration of Soluble VEGFR-3 at Baseline
Time Frame: Baseline (Cycle 1, Day 1)
Population: FA Set
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
pg/mL | 23190 [5480 to 93300] | 23350 [4220 to 413600]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Test type: Superiority or Other; p = 0.9807, Wilcoxon Rank Sum Test — 2-sided normal approximated p-value

67. Secondary Outcome: Plasma Concentration of Soluble KIT (sKIT) at Baseline
Time Frame: Baseline (Cycle 1, Day 1)
Population: FA Set
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Sunitinib + Erlotinib | Erlotinib + Placebo
Number analyzed (Participants) | 65 | 67
pg/mL | 49520 [16870 to 84480] | 47242.50 [21620 to 117900]
Statistical Analysis 1: Comparison: Sunitinib + Erlotinib vs Erlotinib + Placebo; Test type: Superiority or Other; p = 0.3945, Wilcoxon Rank Sum Test — 2-sided normal approximated p-value

ADVERSE EVENTS:
Description: Total number (#) of participants affected/at risk = number of participants with data for summary/number of participants who received at least 1 dose of study treatment
Arm/Group | Sunitinib + Erlotinib (Original Lead-In) | Sunitinib + Erlotinib (Amended Lead-in) | Sunitinib + Erlotinib | Erlotinib + Placebo
Serious Adverse Events (participants affected / at risk) | 5/13 | 7/17 | 29/64 | 28/64
Other Adverse Events (participants affected / at risk) | 13/13 | 15/17 | 60/64 | 61/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib + Erlotinib (Original Lead-In) (N=13) | Sunitinib + Erlotinib (Amended Lead-in) (N=17) | Sunitinib + Erlotinib (N=64) | Erlotinib + Placebo (N=64)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 5 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Femoral hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 4
Asthenia (General disorders) | 0 | 1 | 0 | 1
Disease progression (General disorders) | 1 | 2 | 8 | 8
Fatigue (General disorders) | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Thrombosis in device (General disorders) | 0 | 0 | 0 | 1
Ulcer haemorrhage (General disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 3
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Diabetic hyperosmolar coma (Nervous system disorders) | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 0 | 0 | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Ischaemia (Vascular disorders) | 0 | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib + Erlotinib (Original Lead-In) (N=13) | Sunitinib + Erlotinib (Amended Lead-in) (N=17) | Sunitinib + Erlotinib (N=64) | Erlotinib + Placebo (N=64)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 7 | 4
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 6 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 8 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1
Cyanosis (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 3
Vision blurred (Eye disorders) | 1 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 4 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 7 | 4
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3 | 3 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 9 | 9
Diarrhoea (Gastrointestinal disorders) | 10 | 9 | 37 | 22
Duodenogastric reflux (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 4 | 6
Flatulence (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 1 | 22 | 15
Oral pain (Gastrointestinal disorders) | 2 | 0 | 6 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 5 | 4
Vomiting (Gastrointestinal disorders) | 3 | 2 | 13 | 14
Asthenia (General disorders) | 3 | 0 | 2 | 3
Chest discomfort (General disorders) | 2 | 0 | 1 | 1
Chest pain (General disorders) | 1 | 0 | 2 | 7
Chills (General disorders) | 1 | 0 | 2 | 2
Fatigue (General disorders) | 8 | 2 | 29 | 33
Mucosal inflammation (General disorders) | 1 | 0 | 12 | 7
Oedema peripheral (General disorders) | 2 | 1 | 3 | 4
Pain (General disorders) | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 4 | 1 | 3 | 6
Suprapubic pain (General disorders) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 1 | 1
Infection (Infections and infestations) | 2 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 4
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 2 | 0 | 2 | 3
Pneumonia (Infections and infestations) | 1 | 0 | 3 | 3
Respiratory tract infection (Infections and infestations) | 0 | 1 | 2 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 6 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 1
Blood creatinine increased (Investigations) | 2 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 2 | 3
Platelet count decreased (Investigations) | 1 | 0 | 1 | 0
Vitamin B12 decreased (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 10 | 6
White blood cell count decreased (Investigations) | 2 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 1 | 24 | 20
Dehydration (Metabolism and nutrition disorders) | 5 | 2 | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 6 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5 | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 5 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 7 | 2
Ageusia (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 2 | 2
Dysgeusia (Nervous system disorders) | 4 | 1 | 12 | 6
Headache (Nervous system disorders) | 1 | 0 | 3 | 2
Paraesthesia (Nervous system disorders) | 1 | 0 | 3 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 2 | 2
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 1 | 1
Depression (Psychiatric disorders) | 1 | 0 | 1 | 2
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 5
Dysuria (Renal and urinary disorders) | 1 | 1 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 13 | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 9 | 17
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 4 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5 | 4
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 6 | 0 | 7 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 6
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 3 | 6 | 12
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 20 | 17
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 7
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 5 | 2
Plantar erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 9 | 15
Rash (Skin and subcutaneous tissue disorders) | 6 | 7 | 27 | 19
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 7 | 4
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0
Hypertension (Vascular disorders) | 1 | 4 | 5 | 1
Hypotension (Vascular disorders) | 1 | 0 | 3 | 1
Vena cava thrombosis (Vascular disorders) | 1 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 2
Blepharitis (Eye disorders) | 0 | 0 | 0 | 2
Conjunctivitis (Eye disorders) | 0 | 0 | 3 | 3
Eye irritation (Eye disorders) | 0 | 0 | 1 | 1
Eye pain (Eye disorders) | 0 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 1 | 0
Keratitis (Eye disorders) | 0 | 0 | 1 | 2
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingival disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mouth cyst (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 1
Facial pain (General disorders) | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 1
Localised oedema (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0
Mucous membrane disorder (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 0 | 1
Thrombosis in device (General disorders) | 0 | 0 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 2 | 0
Abscess (Infections and infestations) | 0 | 0 | 1 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0
Conjunctivitis infective (Infections and infestations) | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 2 | 2
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Lip infection (Infections and infestations) | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0
Oral pustule (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia primary atypical (Infections and infestations) | 0 | 0 | 0 | 1
Pulmonary mycosis (Infections and infestations) | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory moniliasis (Infections and infestations) | 0 | 0 | 0 | 1
Superinfection (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 3 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Heat stroke (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0
Granulocyte count decreased (Investigations) | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 2
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 3
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Hypertrophic osteoarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 0 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Spinal cord oedema (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 3 | 1
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1
Nervousness (Psychiatric disorders) | 0 | 0 | 1 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 2 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Haemoglobinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Peyronie's disease (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Alveolar proteinosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Yellow skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 2
Peripheral coldness (Vascular disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Due to rounding some percentages will not equal 100%

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.